CLINICAL TRIAL: NCT02447952
Title: An Exploratory Study to Investigate the Use of Biotelemetry to Identify Markers of Disease Progression in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Exploratory Study of Biotelemetry in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201283
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2017-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Biotelemetry
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot and Core Study Phase (Experimental): During Pilot phase,subjects will attend clinic at least once to perform a series of set reference tasks while wearing the accelerometer and electrode. Subjects will also continuously wear the accelerometer and electrode in their routine home-life setting for approximately 3 days after the clinic visit (home monitoring). During 48 week Core Study, subjects will attend 5 clinic visits to perform gold standard measures of function (ALS Functional Rating Scale-Revised and Forced Vital Capacity) and perform a series of set reference tasks while wearing the accelerometer and electrode. Subjects will also continuously wear the accelerometer and electrode in their routine home-life setting for approximately 3 days after the clinic visits (home monitoring). In between clinic visits, subjects will attach the accelerometer and electrode and wear it for approximately 3 days in their home. A telephone contact with the subject will be made by the site at the end of each 3-day home monitoring period
  Interventions: Device: Faros Sensor (FS) and LifeInsight Hub; Device: Fast Fix electrode patch; Procedure: Quantitative Measure of Speech (Core Phase Only)

INTERVENTIONS:
Device: Faros Sensor (FS) and LifeInsight Hub — Each subject will be issued one FS and a MAT LifeInsight Hub for use during the study. At each clinic visit in the Pilot and Core Study Phases, the Faros sensor will be placed on the subject just prior to the defined reference tasks and will be worn on the subject's sternum during completion of the tasks. The morning after the clinic visit, the subject will re-attach the sensor and wear it for approximately 3 days. In between visits during the Core Study Phase the subject will wear the FS every month for approximately 3 days to enable data collection on a monthly basis over the 48 week study period. Movement/physical activity data will be collected by the FS throughout the study.
Device: Fast Fix electrode patch — The Fast Fix electrode patch will be worn with the FS on the subject's sternum according to the same schedule as the FS. The Fast Fix electrode patch will be replaced by the subject on a daily basis during the 3 day monitoring period. Subjects will be provided instructions on how to operate and wear the Fast Fix electrode patch.
Procedure: Quantitative Measure of Speech (Core Phase Only) — Subjects will follow simple prompts on a computer screen instructing them to say a series of vowels, words, and paragraphs which will be recorded using a high definition digital microphone and stored securely on a laptop. The speech waveform data will be sent via secure method to GSK/MAT for processing.

SUMMARY:
Study 201283 is an exploratory, non-controlled, non-drug study in Amyotrophic Lateral Sclerosis (ALS) subjects. This study is being conducted as the first step for developing new meaningful measure(s) which might prove to be more effective than existing measures for monitoring clinical function and disease course in ALS. The objective of this study is to test novel measures of movement/physical activity, heart rate and speech and explore how they measure disease progression by evaluating their relationship to gold standard measures of function. This study will be conducted in two phases. A variable length Pilot Phase to test biotelemetry instruments and algorithms reliability and ease of use/acceptance. Approximately 5 subjects will have at least 1 clinic visit to perform a series of set reference tasks while wearing the accelerometer and electrode. Subjects will also continuously wear the accelerometer and electrode in their routine home-life setting for approximately 3 days after the clinic visit (i.e., home monitoring). Subjects in the Pilot Phase will continue in the study and participate in the Core Study Phase. A 48 week Core Study Phase will be conducted to evaluate how measures of movement/physical activity, speech and Heart Rate Variability (HRV) relate to ALS disease progression. During this phase, a maximum of 25 subjects will be enrolled. Subjects will attend 5 clinic visits to perform gold standard measures of function and perform a series of set reference tasks while wearing the accelerometer and electrode. In between clinic visits, every month subjects will attach the accelerometer and electrode and wear it for approximately 3 days in their home. A telephone contact with the subject will be made by the site at the end of each 3-day home monitoring period.

All third party trademark rights are the rights of their respective owners.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years of age, inclusive, at the time of signing the informed consent.
* Diagnosed with ALS by a neurologist with expertise in ALS. For subjects with bulbar onset there must be objective limb involvement of at least one limb.
* Diagnosed with ALS within 18 months of symptom onset.
* Subjects must be ambulatory (i.e., must not be confined to a wheelchair).
* Male and female subjects.
* Capable of giving signed (or verbal consent or assent where applicable) informed consent as described in Protocol which includes compliance with the requirements and restrictions listed in the consent form and in protocol.
* Capable and willing to comply with the requirements of the protocol (either by themselves or with assistance).

Exclusion Criteria:

* Neurological (other than the subject's ALS) or non-neurological co-morbidities (e.g. joint disease, respiratory disease) which limit mobility.
* Clinically significant cognitive impairment in the opinion of the investigator.
* Regionally restricted forms of ALS, or other atypical variants: Isolated corticobulbar pattern of ALS with normal ambulation; Flail arm syndrome; Primary lateral sclerosis; Signs of chronic partial denervation restricted to a single limb; ALS parkinsonism dementia complex
* Subjects requiring mechanical ventilation (non-invasive ventilation for sleep apnoea is allowed).
* Historical or current evidence of clinically significant uncontrolled disease which, in the opinion of the investigator, would put the safety of the subject at risk through participation or impact the study assessments or endpoints.
* Presence of an active implantable cardiac medical device (e.g., pacemaker or implantable cardioverter-defibrillator) or at a high risk for needing external defibrillation.
* History of skin hypersensitivity to adhesives.
* Current participation in a clinical trial which in the opinion of the investigator and GSK medical monitor might impact the objectives of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an exploratory, non-controlled, non-drug study in participants with amyotrophic lateral sclerosis (ALS). The study enrolled participants using two sites based in the United Kingdom
Pre-assignment Details: Of total 25 screened participants, 5 participants were included in pilot phase of which 2 completed and entered core study phase with other 23 participants.
Groups:
- Mega Faros Device + Fast Fix: In variable length Pilot Phase participants visited clinic to perform a series of set reference tasks while wearing the accelerometer (Faros device) and electrode (fast fix). Participants continuously wore the accelerometer and electrode in their routine home-life setting for approximately 3 days after the clinic visit (home monitoring). Participants in the Pilot Phase continued to participate in the Core Study Phase. A 48 week Core Study Phase was conducted to evaluate how measures of movement/physical activity, speech and Heart Rate Variability (HRV) relate to ALS disease progression. Participants attended clinic visits to perform gold standard measures of function and perform a series of set reference tasks while wearing the accelerometer and electrode. In between clinic visits, participants attached the accelerometer and electrode and wore it for approximately 3 days in their home.
Period: Overall Study
Arm/Group | Mega Faros Device + Fast Fix
Started | 25
Completed | 18
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 1
  Asian - South East Asian Heritage | 1
  White - White/Caucasian/European Heritage | 23

OUTCOME MEASURES:

1. Primary Outcome: Duration of Day Time Wear Time of the Device
Description: Each participant was provided one accelerometer and electrode (Faros sensor and LifeInsight Hub) through which movement/physical activity data was collected throughout the study. Duration of day time wear time was calculated by adding the durations of the time spent [Active + lying + sedentary not lying] in the day time. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).NA indicates that data could not be calculated as participant number was <=1.
Time Frame: Up to Week 48
Population: Full Analysis Set included all participants with at least one post Baseline measure for the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) and at least one physical activity/movement measure.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Minutes
  Week 0, Day 1, n=24: number analyzed (Participants) | 24
  Week 0, Day 1, n=24 | 718.536 (190.4933)
  Week 0, Day 2, n=24: number analyzed (Participants) | 24
  Week 0, Day 2, n=24 | 730.882 (216.3616)
  Week 0, Day 3, n=23: number analyzed (Participants) | 23
  Week 0, Day 3, n=23 | 653.980 (241.0427)
  Week 0, Day 4, n=12: number analyzed (Participants) | 12
  Week 0, Day 4, n=12 | 207.263 (275.7507)
  Week 0, Day 5, n=2: number analyzed (Participants) | 2
  Week 0, Day 5, n=2 | 342.830 (240.4163)
  Week4, Day 1, n=22: number analyzed (Participants) | 22
  Week4, Day 1, n=22 | 762.680 (228.5267)
  Week4, Day 2, n=22: number analyzed (Participants) | 22
  Week4, Day 2, n=22 | 778.636 (169.6978)
  Week4, Day 3, n=21: number analyzed (Participants) | 21
  Week4, Day 3, n=21 | 605.334 (319.5373)
  Week4, Day 4, n=9: number analyzed (Participants) | 9
  Week4, Day 4, n=9 | 207.092 (293.8405)
  Week4, Day 5, n=5: number analyzed (Participants) | 5
  Week4, Day 5, n=5 | 137.600 (300.5371)
  Week4, Day 6, n=1: number analyzed (Participants) | 1
  Week4, Day 6, n=1 | 657.500 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week4, Day 7, n=1: number analyzed (Participants) | 1
  Week4, Day 7, n=1 | 820.660 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week4, Day 8, n=1: number analyzed (Participants) | 1
  Week4, Day 8, n=1 | 34.000 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week8, Day 1, n=19: number analyzed (Participants) | 19
  Week8, Day 1, n=19 | 647.735 (291.5468)
  Week8, Day 2, n=17: number analyzed (Participants) | 17
  Week8, Day 2, n=17 | 744.028 (158.3890)
  Week8, Day 3, n=17: number analyzed (Participants) | 17
  Week8, Day 3, n=17 | 581.939 (297.5053)
  Week8, Day 4, n=8: number analyzed (Participants) | 8
  Week8, Day 4, n=8 | 94.709 (126.7088)
  Week12,Day 1, n=16: number analyzed (Participants) | 16
  Week12,Day 1, n=16 | 552.668 (315.5227)
  Week12,Day 2, n=16: number analyzed (Participants) | 16
  Week12,Day 2, n=16 | 801.697 (170.8600)
  Week12,Day 3, n=15: number analyzed (Participants) | 15
  Week12,Day 3, n=15 | 563.311 (298.3566)
  Week12,Day 4, n=7: number analyzed (Participants) | 7
  Week12,Day 4, n=7 | 425.336 (266.8420)
  Week12,Day 5, n=1: number analyzed (Participants) | 1
  Week12,Day 5, n=1 | 858.660 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week16,Day 1, n=13: number analyzed (Participants) | 13
  Week16,Day 1, n=13 | 759.399 (129.2502)
  Week16,Day 2, n=13: number analyzed (Participants) | 13
  Week16,Day 2, n=13 | 812.345 (200.5683)
  Week16,Day 3, n=12: number analyzed (Participants) | 12
  Week16,Day 3, n=12 | 631.484 (296.3050)
  Week16,Day 4, n=6: number analyzed (Participants) | 6
  Week16,Day 4, n=6 | 254.500 (336.6649)
  Week20,Day 1, n=14: number analyzed (Participants) | 14
  Week20,Day 1, n=14 | 774.049 (240.7234)
  Week20,Day 2, n=13: number analyzed (Participants) | 13
  Week20,Day 2, n=13 | 648.268 (291.9654)
  Week20,Day 3, n=12: number analyzed (Participants) | 12
  Week20,Day 3, n=12 | 615.277 (239.5376)
  Week20,Day 4, n=4: number analyzed (Participants) | 4
  Week20,Day 4, n=4 | 172.793 (345.3584)
  Week24,Day 1, n=14: number analyzed (Participants) | 14
  Week24,Day 1, n=14 | 505.976 (296.3016)
  Week24,Day 2, n=12: number analyzed (Participants) | 12
  Week24,Day 2, n=12 | 617.599 (299.5749)
  Week24,Day 3, n=11: number analyzed (Participants) | 11
  Week24,Day 3, n=11 | 481.698 (333.5209)
  Week24,Day 4, n=8: number analyzed (Participants) | 8
  Week24,Day 4, n=8 | 306.500 (303.9026)
  Week24,Day 5, n=2: number analyzed (Participants) | 2
  Week24,Day 5, n=2 | 287.000 (184.7953)
  Week28,Day 1, n=10: number analyzed (Participants) | 10
  Week28,Day 1, n=10 | 690.898 (178.9577)
  Week28,Day 2, n=10: number analyzed (Participants) | 10
  Week28,Day 2, n=10 | 722.551 (248.5576)
  Week28,Day 3, n=9: number analyzed (Participants) | 9
  Week28,Day 3, n=9 | 588.464 (359.3972)
  Week28,Day 4, n=6: number analyzed (Participants) | 6
  Week28,Day 4, n=6 | 357.220 (363.2050)
  Week32,Day 1, n=12: number analyzed (Participants) | 12
  Week32,Day 1, n=12 | 575.303 (322.1123)
  Week32,Day 2, n=10: number analyzed (Participants) | 10
  Week32,Day 2, n=10 | 592.866 (345.4597)
  Week32,Day 3, n=9: number analyzed (Participants) | 9
  Week32,Day 3, n=9 | 599.778 (351.8631)
  Week32,Day 4, n=1: number analyzed (Participants) | 1
  Week32,Day 4, n=1 | 32.000 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week36,Day 1, n=12: number analyzed (Participants) | 12
  Week36,Day 1, n=12 | 510.209 (381.7060)
  Week36,Day 2, n=9: number analyzed (Participants) | 9
  Week36,Day 2, n=9 | 507.872 (397.7501)
  Week36,Day 3, n=6: number analyzed (Participants) | 6
  Week36,Day 3, n=6 | 465.583 (340.8965)
  Week36,Day 4, n=4: number analyzed (Participants) | 4
  Week36,Day 4, n=4 | 387.750 (424.1863)
  Week36,Day 5, n=2: number analyzed (Participants) | 2
  Week36,Day 5, n=2 | 516.250 (454.3161)
  Week36,Day 6, n=1: number analyzed (Participants) | 1
  Week36,Day 6, n=1 | 171.840 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week40,Day 1, n=12: number analyzed (Participants) | 12
  Week40,Day 1, n=12 | 722.708 (239.1189)
  Week40,Day 2, n=12: number analyzed (Participants) | 12
  Week40,Day 2, n=12 | 618.555 (326.7927)
  Week40,Day 3, n=11: number analyzed (Participants) | 11
  Week40,Day 3, n=11 | 601.665 (312.9329)
  Week40,Day 4, n=7: number analyzed (Participants) | 7
  Week40,Day 4, n=7 | 290.857 (404.5156)
  Week40,Day 5, n=1: number analyzed (Participants) | 1
  Week40,Day 5, n=1 | 823.500 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week40,Day 6, n=1: number analyzed (Participants) | 1
  Week40,Day 6, n=1 | 444.830 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week44,Day 1, n=12: number analyzed (Participants) | 12
  Week44,Day 1, n=12 | 746.278 (258.7132)
  Week44,Day 2, n=11: number analyzed (Participants) | 11
  Week44,Day 2, n=11 | 646.452 (295.5684)
  Week44,Day 3, n=10: number analyzed (Participants) | 10
  Week44,Day 3, n=10 | 476.783 (355.1196)
  Week44,Day 4, n=4: number analyzed (Participants) | 4
  Week44,Day 4, n=4 | 178.460 (308.3123)
  Week44,Day 5, n=1: number analyzed (Participants) | 1
  Week44,Day 5, n=1 | 146.660 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week48,Day 1, n=13: number analyzed (Participants) | 13
  Week48,Day 1, n=13 | 779.438 (120.7527)
  Week48,Day 2, n=13: number analyzed (Participants) | 13
  Week48,Day 2, n=13 | 692.474 (251.7305)
  Week48,Day 3, n=10: number analyzed (Participants) | 10
  Week48,Day 3, n=10 | 622.015 (243.5040)
  Week48,Day 4, n=5: number analyzed (Participants) | 5
  Week48,Day 4, n=5 | 630.000 (380.2256)

2. Other Pre Specified Outcome: Duration of Night Time Wear Time of the Device
Description: Each participant was provided one accelerometer and electrode (Faros sensor and LifeInsight Hub) through which movement/physical activity data was collected throughout the study. Duration of night time wear time was the calculated as the total of the times spent [Active + day time lying + day time "sedentary not lying"] for the night time. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data could not be calculated as participant number was <=1.
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Minutes
  Week 0, Day 1, n=24: number analyzed (Participants) | 24
  Week 0, Day 1, n=24 | 448.174 (222.1658)
  Week 0, Day 2, n=24: number analyzed (Participants) | 24
  Week 0, Day 2, n=24 | 360.575 (212.4216)
  Week 0, Day 3, n=23: number analyzed (Participants) | 23
  Week 0, Day 3, n=23 | 482.500 (150.8251)
  Week 0, Day 4, n=12: number analyzed (Participants) | 12
  Week 0, Day 4, n=12 | 134.570 (239.8401)
  Week 0, Day 5, n=2: number analyzed (Participants) | 2
  Week 0, Day 5, n=2 | 494.170 (57.9828)
  Week4, Day 1, n=22: number analyzed (Participants) | 22
  Week4, Day 1, n=22 | 487.682 (189.6054)
  Week4, Day 2, n=22: number analyzed (Participants) | 22
  Week4, Day 2, n=22 | 432.273 (209.9463)
  Week4, Day 3, n=21: number analyzed (Participants) | 21
  Week4, Day 3, n=21 | 455.047 (194.3802)
  Week4, Day 4, n=9: number analyzed (Participants) | 9
  Week4, Day 4, n=9 | 107.796 (205.8403)
  Week4, Day 5, n=5: number analyzed (Participants) | 5
  Week4, Day 5, n=5 | 109.400 (241.1904)
  Week4, Day 6, n=1: number analyzed (Participants) | 1
  Week4, Day 6, n=1 | 624.500 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week4, Day 7, n=1: number analyzed (Participants) | 1
  Week4, Day 7, n=1 | 462.340 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week4, Day 8, n=1: number analyzed (Participants) | 1
  Week4, Day 8, n=1 | 0.000 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week8, Day 1, n=19: number analyzed (Participants) | 19
  Week8, Day 1, n=19 | 506.316 (184.6635)
  Week8, Day 2, n=17: number analyzed (Participants) | 17
  Week8, Day 2, n=17 | 477.441 (206.7924)
  Week8, Day 3, n=17: number analyzed (Participants) | 17
  Week8, Day 3, n=17 | 526.825 (207.6252)
  Week8, Day 4, n=8: number analyzed (Participants) | 8
  Week8, Day 4, n=8 | 30.041 (84.9695)
  Week12,Day 1, n=16: number analyzed (Participants) | 16
  Week12,Day 1, n=16 | 255.708 (250.9718)
  Week12,Day 2, n=16: number analyzed (Participants) | 16
  Week12,Day 2, n=16 | 418.489 (149.6411)
  Week12,Day 3, n=15: number analyzed (Participants) | 15
  Week12,Day 3, n=15 | 519.888 (63.0517)
  Week12,Day 4, n=7: number analyzed (Participants) | 7
  Week12,Day 4, n=7 | 568.381 (150.2560)
  Week12,Day 5, n=1: number analyzed (Participants) | 1
  Week12,Day 5, n=1 | 406.340 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week16,Day 1, n=13: number analyzed (Participants) | 13
  Week16,Day 1, n=13 | 513.448 (78.9644)
  Week16,Day 2, n=13: number analyzed (Participants) | 13
  Week16,Day 2, n=13 | 382.038 (185.6318)
  Week16,Day 3, n=12: number analyzed (Participants) | 12
  Week16,Day 3, n=12 | 494.932 (196.5556)
  Week16,Day 4, n=6: number analyzed (Participants) | 6
  Week16,Day 4, n=6 | 96.000 (220.5519)
  Week20,Day 1, n=14: number analyzed (Participants) | 14
  Week20,Day 1, n=14 | 445.811 (170.4490)
  Week20,Day 2, n=13: number analyzed (Participants) | 13
  Week20,Day 2, n=13 | 452.345 (203.3159)
  Week20,Day 3, n=12: number analyzed (Participants) | 12
  Week20,Day 3, n=12 | 498.806 (138.8339)
  Week20,Day 4, n=4: number analyzed (Participants) | 4
  Week20,Day 4, n=4 | 148.458 (172.2844)
  Week24,Day 1, n=14: number analyzed (Participants) | 14
  Week24,Day 1, n=14 | 254.095 (261.1246)
  Week24,Day 2, n=12: number analyzed (Participants) | 12
  Week24,Day 2, n=12 | 398.068 (199.7096)
  Week24,Day 3, n=11: number analyzed (Participants) | 11
  Week24,Day 3, n=11 | 374.121 (214.6214)
  Week24,Day 4, n=8: number analyzed (Participants) | 8
  Week24,Day 4, n=8 | 291.376 (277.4058)
  Week24,Day 5, n=2: number analyzed (Participants) | 2
  Week24,Day 5, n=2 | 476.995 (1.8880)
  Week28,Day 1, n=10: number analyzed (Participants) | 10
  Week28,Day 1, n=10 | 497.701 (242.6652)
  Week28,Day 2, n=10: number analyzed (Participants) | 10
  Week28,Day 2, n=10 | 483.950 (195.5384)
  Week28,Day 3, n=9: number analyzed (Participants) | 9
  Week28,Day 3, n=9 | 543.759 (270.4945)
  Week28,Day 4, n=6: number analyzed (Participants) | 6
  Week28,Day 4, n=6 | 286.778 (327.2635)
  Week32,Day 1, n=12: number analyzed (Participants) | 12
  Week32,Day 1, n=12 | 510.447 (218.5192)
  Week32,Day 2, n=10: number analyzed (Participants) | 10
  Week32,Day 2, n=10 | 460.233 (209.0824)
  Week32,Day 3, n=9: number analyzed (Participants) | 9
  Week32,Day 3, n=9 | 433.778 (256.9437)
  Week32,Day 4, n=1: number analyzed (Participants) | 1
  Week32,Day 4, n=1 | 0.000 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week36,Day 1, n=12: number analyzed (Participants) | 12
  Week36,Day 1, n=12 | 189.124 (199.2290)
  Week36,Day 2, n=9: number analyzed (Participants) | 9
  Week36,Day 2, n=9 | 263.352 (236.3438)
  Week36,Day 3, n=6: number analyzed (Participants) | 6
  Week36,Day 3, n=6 | 380.748 (298.7767)
  Week36,Day 4, n=4: number analyzed (Participants) | 4
  Week36,Day 4, n=4 | 358.503 (280.5689)
  Week36,Day 5, n=2: number analyzed (Participants) | 2
  Week36,Day 5, n=2 | 201.250 (284.6105)
  Week36,Day 6, n=1: number analyzed (Participants) | 1
  Week36,Day 6, n=1 | 505.170 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week40,Day 1, n=12: number analyzed (Participants) | 12
  Week40,Day 1, n=12 | 375.043 (192.0867)
  Week40,Day 2, n=12: number analyzed (Participants) | 12
  Week40,Day 2, n=12 | 442.528 (179.2818)
  Week40,Day 3, n=11: number analyzed (Participants) | 11
  Week40,Day 3, n=11 | 419.334 (215.0470)
  Week40,Day 4, n=7: number analyzed (Participants) | 7
  Week40,Day 4, n=7 | 121.573 (172.7203)
  Week40,Day 5, n=1: number analyzed (Participants) | 1
  Week40,Day 5, n=1 | 522.500 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week40,Day 6, n=1: number analyzed (Participants) | 1
  Week40,Day 6, n=1 | 163.170 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week44,Day 1, n=12: number analyzed (Participants) | 12
  Week44,Day 1, n=12 | 393.140 (192.6969)
  Week44,Day 2, n=11: number analyzed (Participants) | 11
  Week44,Day 2, n=11 | 362.275 (208.9128)
  Week44,Day 3, n=10: number analyzed (Participants) | 10
  Week44,Day 3, n=10 | 382.018 (201.1957)
  Week44,Day 4, n=4: number analyzed (Participants) | 4
  Week44,Day 4, n=4 | 111.543 (223.0850)
  Week44,Day 5, n=1: number analyzed (Participants) | 1
  Week44,Day 5, n=1 | 277.330 (NA) — NA indicates that data could not be calculated as participant number was <=1.
  Week48,Day 1, n=13: number analyzed (Participants) | 13
  Week48,Day 1, n=13 | 439.486 (153.3470)
  Week48,Day 2, n=13: number analyzed (Participants) | 13
  Week48,Day 2, n=13 | 381.988 (192.9540)
  Week48,Day 3, n=10: number analyzed (Participants) | 10
  Week48,Day 3, n=10 | 299.985 (146.9104)
  Week48,Day 4, n=5: number analyzed (Participants) | 5
  Week48,Day 4, n=5 | 81.400 (182.0159)

3. Other Pre Specified Outcome: Average Time Spent Active
Description: Number of minutes spent active per day and night over the 24-hour recording periods; averaged for each time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Minutes
  Day time, Week 0, n=24: number analyzed (Participants) | 24
  Day time, Week 0, n=24 | 34.420 (29.3837)
  Day time, Week 4, n=22: number analyzed (Participants) | 22
  Day time, Week 4, n=22 | 32.233 (33.1012)
  Day time, Week 8, n=19: number analyzed (Participants) | 19
  Day time, Week 8, n=19 | 24.319 (25.5092)
  Day time, Week 12, n=16: number analyzed (Participants) | 16
  Day time, Week 12, n=16 | 23.904 (17.2952)
  Day time, Week 16, n=13: number analyzed (Participants) | 13
  Day time, Week 16, n=13 | 25.863 (23.2673)
  Day time, Week 20, n=14: number analyzed (Participants) | 14
  Day time, Week 20, n=14 | 18.931 (18.3595)
  Day time, Week 24, n=14: number analyzed (Participants) | 14
  Day time, Week 24, n=14 | 12.137 (10.8409)
  Day time, Week 28, n=10: number analyzed (Participants) | 10
  Day time, Week 28, n=10 | 19.856 (29.0562)
  Day time, Week 32, n=12: number analyzed (Participants) | 12
  Day time, Week 32, n=12 | 11.873 (15.0988)
  Day time, Week 36, n=12: number analyzed (Participants) | 12
  Day time, Week 36, n=12 | 14.118 (19.7452)
  Day time, Week 40, n=12: number analyzed (Participants) | 12
  Day time, Week 40, n=12 | 14.563 (18.7912)
  Day time, Week 44, n=12: number analyzed (Participants) | 12
  Day time, Week 44, n=12 | 20.210 (26.0361)
  Day time, Week 48, n=13: number analyzed (Participants) | 13
  Day time, Week 48, n=13 | 23.578 (29.0419)
  Night time, Week 0, n=24: number analyzed (Participants) | 24
  Night time, Week 0, n=24 | 1.136 (1.5427)
  Night time, Week 4, n=22: number analyzed (Participants) | 22
  Night time, Week 4, n=22 | 0.570 (0.6817)
  Night time, Week 8, n=19: number analyzed (Participants) | 19
  Night time, Week 8, n=19 | 2.375 (5.7540)
  Night time, Week 12, n=16: number analyzed (Participants) | 16
  Night time, Week 12, n=16 | 0.484 (0.5404)
  Night time, Week 16, n=13: number analyzed (Participants) | 13
  Night time, Week 16, n=13 | 0.449 (0.4684)
  Night time, Week 20, n=14: number analyzed (Participants) | 14
  Night time, Week 20, n=14 | 0.418 (0.5315)
  Night time, Week 24, n=14: number analyzed (Participants) | 14
  Night time, Week 24, n=14 | 0.387 (0.2715)
  Night time, Week 28, n=10: number analyzed (Participants) | 10
  Night time, Week 28, n=10 | 1.432 (3.0455)
  Night time, Week 32, n=12: number analyzed (Participants) | 12
  Night time, Week 32, n=12 | 0.668 (1.5814)
  Night time, Week 36, n=12: number analyzed (Participants) | 12
  Night time, Week 36, n=12 | 0.414 (0.3682)
  Night time, Week 40, n=12: number analyzed (Participants) | 12
  Night time, Week 40, n=12 | 0.268 (0.3272)
  Night time, Week 44, n=12: number analyzed (Participants) | 12
  Night time, Week 44, n=12 | 0.390 (0.7308)
  Night time, Week 48, n=13: number analyzed (Participants) | 13
  Night time, Week 48, n=13 | 0.518 (0.8014)

4. Other Pre Specified Outcome: Average Time Spent 'Sedentary Not Lying'
Description: Number of minutes spent 'sedentary not lying' per day and night for 24-hour recording period; averaged for each time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Minutes
  Day time, Week 0, n=24: number analyzed (Participants) | 24
  Day time, Week 0, n=24 | 523.191 (113.3016)
  Day time, Week 4, n=22: number analyzed (Participants) | 22
  Day time, Week 4, n=22 | 524.120 (182.7753)
  Day time, Week 8, n=19: number analyzed (Participants) | 19
  Day time, Week 8, n=19 | 428.359 (210.1894)
  Day time, Week 12, n=16: number analyzed (Participants) | 16
  Day time, Week 12, n=16 | 509.634 (105.3263)
  Day time, Week 16, n=13: number analyzed (Participants) | 13
  Day time, Week 16, n=13 | 561.923 (100.3003)
  Day time, Week 20, n=14: number analyzed (Participants) | 14
  Day time, Week 20, n=14 | 489.921 (202.2926)
  Day time, Week 24, n=14: number analyzed (Participants) | 14
  Day time, Week 24, n=14 | 376.117 (222.6009)
  Day time, Week 28, n=10: number analyzed (Participants) | 10
  Day time, Week 28, n=10 | 472.238 (215.7768)
  Day time, Week 32, n=12: number analyzed (Participants) | 12
  Day time, Week 32, n=12 | 420.709 (259.0856)
  Day time, Week 36, n=12: number analyzed (Participants) | 12
  Day time, Week 36, n=12 | 376.686 (233.1990)
  Day time, Week 40, n=12: number analyzed (Participants) | 12
  Day time, Week 40, n=12 | 465.879 (181.5005)
  Day time, Week 44, n=12: number analyzed (Participants) | 12
  Day time, Week 44, n=12 | 440.376 (198.2569)
  Day time, Week 48, n=13: number analyzed (Participants) | 13
  Day time, Week 48, n=13 | 509.536 (171.1560)
  Night time, Week 0, n=24: number analyzed (Participants) | 24
  Night time, Week 0, n=24 | 15.522 (28.5337)
  Night time, Week 4, n=22: number analyzed (Participants) | 22
  Night time, Week 4, n=22 | 10.561 (12.5485)
  Night time, Week 8, n=19: number analyzed (Participants) | 19
  Night time, Week 8, n=19 | 8.441 (5.8601)
  Night time, Week 12, n=16: number analyzed (Participants) | 16
  Night time, Week 12, n=16 | 7.968 (4.8657)
  Night time, Week 16, n=13: number analyzed (Participants) | 13
  Night time, Week 16, n=13 | 8.855 (5.1855)
  Night time, Week 20, n=14: number analyzed (Participants) | 14
  Night time, Week 20, n=14 | 9.239 (6.9942)
  Night time, Week 24, n=14: number analyzed (Participants) | 14
  Night time, Week 24, n=14 | 7.274 (6.5610)
  Night time, Week 28, n=10: number analyzed (Participants) | 10
  Night time, Week 28, n=10 | 17.488 (15.1698)
  Night time, Week 32, n=12: number analyzed (Participants) | 12
  Night time, Week 32, n=12 | 12.930 (14.8779)
  Night time, Week 36, n=12: number analyzed (Participants) | 12
  Night time, Week 36, n=12 | 3.545 (3.5805)
  Night time, Week 40, n=12: number analyzed (Participants) | 12
  Night time, Week 40, n=12 | 8.932 (5.0236)
  Night time, Week 44, n=12: number analyzed (Participants) | 12
  Night time, Week 44, n=12 | 6.321 (4.5166)
  Night time, Week 48, n=13: number analyzed (Participants) | 13
  Night time, Week 48, n=13 | 7.602 (7.4373)

5. Other Pre Specified Outcome: Average Time Spent Lying
Description: Number of minutes spent lying per day and night over the 24-hour recording periods; averaged for each time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Minutes
  Day time, Week 0, n=24: number analyzed (Participants) | 24
  Day time, Week 0, n=24 | 79.027 (59.8512)
  Day time, Week 4, n=22: number analyzed (Participants) | 22
  Day time, Week 4, n=22 | 79.996 (67.1924)
  Day time, Week 8, n=19: number analyzed (Participants) | 19
  Day time, Week 8, n=19 | 90.324 (80.8799)
  Day time, Week 12, n=16: number analyzed (Participants) | 16
  Day time, Week 12, n=16 | 82.146 (59.7457)
  Day time, Week 16, n=13: number analyzed (Participants) | 13
  Day time, Week 16, n=13 | 87.271 (75.4731)
  Day time, Week 20, n=14: number analyzed (Participants) | 14
  Day time, Week 20, n=14 | 89.648 (90.8020)
  Day time, Week 24, n=14: number analyzed (Participants) | 14
  Day time, Week 24, n=14 | 82.979 (89.4852)
  Day time, Week 28, n=10: number analyzed (Participants) | 10
  Day time, Week 28, n=10 | 136.170 (127.2225)
  Day time, Week 32, n=12: number analyzed (Participants) | 12
  Day time, Week 32, n=12 | 99.760 (118.3536)
  Day time, Week 36, n=12: number analyzed (Participants) | 12
  Day time, Week 36, n=12 | 50.278 (48.7456)
  Day time, Week 40, n=12: number analyzed (Participants) | 12
  Day time, Week 40, n=12 | 103.749 (133.3234)
  Day time, Week 44, n=12: number analyzed (Participants) | 12
  Day time, Week 44, n=12 | 71.757 (73.5817)
  Day time, Week 48, n=13: number analyzed (Participants) | 13
  Day time, Week 48, n=13 | 141.575 (140.1450)
  Night time, Week 0, n=24: number analyzed (Participants) | 24
  Night time, Week 0, n=24 | 384.886 (135.8136)
  Night time, Week 4, n=22: number analyzed (Participants) | 22
  Night time, Week 4, n=22 | 384.879 (97.8424)
  Night time, Week 8, n=19: number analyzed (Participants) | 19
  Night time, Week 8, n=19 | 411.110 (157.8820)
  Night time, Week 12, n=16: number analyzed (Participants) | 16
  Night time, Week 12, n=16 | 417.943 (71.9066)
  Night time, Week 16, n=13: number analyzed (Participants) | 13
  Night time, Week 16, n=13 | 413.721 (129.3161)
  Night time, Week 20, n=14: number analyzed (Participants) | 14
  Night time, Week 20, n=14 | 407.060 (175.2092)
  Night time, Week 24, n=14: number analyzed (Participants) | 14
  Night time, Week 24, n=14 | 318.155 (112.8749)
  Night time, Week 28, n=10: number analyzed (Participants) | 10
  Night time, Week 28, n=10 | 454.137 (184.2617)
  Night time, Week 32, n=12: number analyzed (Participants) | 12
  Night time, Week 32, n=12 | 412.196 (170.4452)
  Night time, Week 36, n=12: number analyzed (Participants) | 12
  Night time, Week 36, n=12 | 217.884 (181.3682)
  Night time, Week 40, n=12: number analyzed (Participants) | 12
  Night time, Week 40, n=12 | 355.222 (104.8680)
  Night time, Week 44, n=12: number analyzed (Participants) | 12
  Night time, Week 44, n=12 | 319.022 (155.2519)
  Night time, Week 48, n=13: number analyzed (Participants) | 13
  Night time, Week 48, n=13 | 333.358 (154.9236)

6. Other Pre Specified Outcome: Average Time Spent Sedentary.
Description: Number of minutes spent sedentary [time spent lying + time spent sedentary not lying] per day and night over the 24-hour recording periods; averaged for each time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Minutes
  Day time, Week 0, n=24: number analyzed (Participants) | 24
  Day time, Week 0, n=24 | 602.219 (131.7430)
  Day time, Week 4, n=22: number analyzed (Participants) | 22
  Day time, Week 4, n=22 | 604.116 (165.0799)
  Day time, Week 8, n=19: number analyzed (Participants) | 19
  Day time, Week 8, n=19 | 518.684 (234.6306)
  Day time, Week 12, n=16: number analyzed (Participants) | 16
  Day time, Week 12, n=16 | 591.779 (118.3797)
  Day time, Week 16, n=13: number analyzed (Participants) | 13
  Day time, Week 16, n=13 | 649.195 (117.2721)
  Day time, Week 20, n=14: number analyzed (Participants) | 14
  Day time, Week 20, n=14 | 579.571 (213.9093)
  Day time, Week 24, n=14: number analyzed (Participants) | 14
  Day time, Week 24, n=14 | 459.096 (233.1413)
  Day time, Week 28, n=10: number analyzed (Participants) | 10
  Day time, Week 28, n=10 | 608.409 (141.5444)
  Day time, Week 32, n=12: number analyzed (Participants) | 12
  Day time, Week 32, n=12 | 520.468 (285.7109)
  Day time, Week 36, n=12: number analyzed (Participants) | 12
  Day time, Week 36, n=12 | 426.962 (250.2390)
  Day time, Week 40, n=12: number analyzed (Participants) | 12
  Day time, Week 40, n=12 | 569.629 (171.5586)
  Day time, Week 44, n=12: number analyzed (Participants) | 12
  Day time, Week 44, n=12 | 512.132 (203.0705)
  Day time, Week 48, n=13: number analyzed (Participants) | 13
  Day time, Week 48, n=13 | 651.109 (156.3296)
  Night time, Week 0, n=24: number analyzed (Participants) | 24
  Night time, Week 0, n=24 | 400.408 (132.3420)
  Night time, Week 4, n=22: number analyzed (Participants) | 22
  Night time, Week 4, n=22 | 395.438 (100.9179)
  Night time, Week 8, n=19: number analyzed (Participants) | 19
  Night time, Week 8, n=19 | 419.549 (162.0795)
  Night time, Week 12, n=16: number analyzed (Participants) | 16
  Night time, Week 12, n=16 | 425.909 (69.7741)
  Night time, Week 16, n=13: number analyzed (Participants) | 13
  Night time, Week 16, n=13 | 422.574 (132.3307)
  Night time, Week 20, n=14: number analyzed (Participants) | 14
  Night time, Week 20, n=14 | 416.299 (179.9825)
  Night time, Week 24, n=14: number analyzed (Participants) | 14
  Night time, Week 24, n=14 | 325.427 (114.9446)
  Night time, Week 28, n=10: number analyzed (Participants) | 10
  Night time, Week 28, n=10 | 471.626 (196.1417)
  Night time, Week 32, n=12: number analyzed (Participants) | 12
  Night time, Week 32, n=12 | 425.125 (178.8053)
  Night time, Week 36, n=12: number analyzed (Participants) | 12
  Night time, Week 36, n=12 | 221.430 (184.4017)
  Night time, Week 40, n=12: number analyzed (Participants) | 12
  Night time, Week 40, n=12 | 364.152 (105.2901)
  Night time, Week 44, n=12: number analyzed (Participants) | 12
  Night time, Week 44, n=12 | 325.343 (156.8669)
  Night time, Week 48, n=13: number analyzed (Participants) | 13
  Night time, Week 48, n=13 | 340.960 (157.6860)

7. Other Pre Specified Outcome: Time Spent With Sensor Off
Description: Sensor off time includes the time that the sensor was either switched off or the participant was not wearing it (or both). This outcome measure was planned but not performed.
Time Frame: Up to Week 48
Population: Full Analysis Set
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Total Activity Count
Description: Total activity count for the day time and night time for the 24-hour recording periods; averaged for each time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Count of activity
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Count of activity
  Day time, Week 0, n=24: number analyzed (Participants) | 24
  Day time, Week 0, n=24 | 3336.550 (2654.406)
  Day time, Week 4, n=22: number analyzed (Participants) | 22
  Day time, Week 4, n=22 | 2903.633 (3059.200)
  Day time, Week 8, n=17: number analyzed (Participants) | 17
  Day time, Week 8, n=17 | 4244.521 (6314.828)
  Day time, Week 12, n=16: number analyzed (Participants) | 16
  Day time, Week 12, n=16 | 2076.129 (1338.276)
  Day time, Week 16, n=13: number analyzed (Participants) | 13
  Day time, Week 16, n=13 | 2216.162 (1732.185)
  Day time, Week 20, n=14: number analyzed (Participants) | 14
  Day time, Week 20, n=14 | 1858.116 (1504.067)
  Day time, Week 24, n=13: number analyzed (Participants) | 13
  Day time, Week 24, n=13 | 1114.152 (683.2223)
  Day time, Week 28, n=10: number analyzed (Participants) | 10
  Day time, Week 28, n=10 | 1468.741 (1559.431)
  Day time, Week 32, n=12: number analyzed (Participants) | 12
  Day time, Week 32, n=12 | 1247.969 (1015.319)
  Day time, Week 36, n=12: number analyzed (Participants) | 12
  Day time, Week 36, n=12 | 1675.754 (1979.210)
  Day time, Week 40, n=12: number analyzed (Participants) | 12
  Day time, Week 40, n=12 | 1542.138 (1421.696)
  Day time, Week 44, n=12: number analyzed (Participants) | 12
  Day time, Week 44, n=12 | 2252.325 (1923.793)
  Day time, Week 48, n=13: number analyzed (Participants) | 13
  Day time, Week 48, n=13 | 1972.506 (2209.802)
  Night time, Week 0, n=24: number analyzed (Participants) | 24
  Night time, Week 0, n=24 | 357.865 (293.7938)
  Night time, Week 4, n=22: number analyzed (Participants) | 22
  Night time, Week 4, n=22 | 265.096 (102.7897)
  Night time, Week 8, n=13: number analyzed (Participants) | 13
  Night time, Week 8, n=13 | 652.108 (1445.624)
  Night time, Week 12, n=16: number analyzed (Participants) | 16
  Night time, Week 12, n=16 | 234.854 (68.8019)
  Night time, Week 16, n=13: number analyzed (Participants) | 13
  Night time, Week 16, n=13 | 254.238 (46.4883)
  Night time, Week 20, n=14: number analyzed (Participants) | 14
  Night time, Week 20, n=14 | 241.504 (68.9048)
  Night time, Week 24, n=14: number analyzed (Participants) | 14
  Night time, Week 24, n=14 | 249.504 (165.5673)
  Night time, Week 28, n=10: number analyzed (Participants) | 10
  Night time, Week 28, n=10 | 328.374 (222.3131)
  Night time, Week 32, n=12: number analyzed (Participants) | 12
  Night time, Week 32, n=12 | 271.988 (189.5221)
  Night time, Week 36, n=10: number analyzed (Participants) | 10
  Night time, Week 36, n=10 | 211.270 (101.4570)
  Night time, Week 40, n=12: number analyzed (Participants) | 12
  Night time, Week 40, n=12 | 212.134 (68.5433)
  Night time, Week 44, n=11: number analyzed (Participants) | 11
  Night time, Week 44, n=11 | 232.571 (117.1910)
  Night time, Week 48, n=13: number analyzed (Participants) | 13
  Night time, Week 48, n=13 | 224.375 (110.9312)

9. Other Pre Specified Outcome: Maximum Activity Count in a 24 Hour Period
Description: Maximum activity count for the day time and night time for the 24-hour recording periods; averaged for each time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Count of activity
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Count of activity
  Day time, Week 0, n=24: number analyzed (Participants) | 24
  Day time, Week 0, n=24 | 2803.906 (2819.342)
  Day time, Week 4, n=22: number analyzed (Participants) | 22
  Day time, Week 4, n=22 | 1915.344 (1787.325)
  Day time, Week 8, n=17: number analyzed (Participants) | 17
  Day time, Week 8, n=17 | 3520.196 (6145.555)
  Day time, Week 12, n=16: number analyzed (Participants) | 16
  Day time, Week 12, n=16 | 2004.569 (1341.035)
  Day time, Week 16, n=13: number analyzed (Participants) | 13
  Day time, Week 16, n=13 | 2337.092 (2537.966)
  Day time, Week 20, n=14: number analyzed (Participants) | 14
  Day time, Week 20, n=14 | 1923.578 (1690.000)
  Day time, Week 24, n=13: number analyzed (Participants) | 13
  Day time, Week 24, n=13 | 1050.409 (831.3745)
  Day time, Week 28, n=10: number analyzed (Participants) | 10
  Day time, Week 28, n=10 | 960.596 (667.9179)
  Day time, Week 32, n=12: number analyzed (Participants) | 12
  Day time, Week 32, n=12 | 815.954 (772.5387)
  Day time, Week 36, n=12: number analyzed (Participants) | 12
  Day time, Week 36, n=12 | 1238.367 (1121.657)
  Day time, Week 40, n=12: number analyzed (Participants) | 12
  Day time, Week 40, n=12 | 897.363 (785.0252)
  Day time, Week 44, n=12: number analyzed (Participants) | 12
  Day time, Week 44, n=12 | 1940.100 (2346.428)
  Day time, Week 48, n=13: number analyzed (Participants) | 13
  Day time, Week 48, n=13 | 1647.037 (1645.568)
  Night time, Week 0, n=24: number analyzed (Participants) | 24
  Night time, Week 0, n=24 | 657.385 (823.5054)
  Night time, Week 4, n=22: number analyzed (Participants) | 22
  Night time, Week 4, n=22 | 511.867 (599.0219)
  Night time, Week 8, n=19: number analyzed (Participants) | 19
  Night time, Week 8, n=19 | 676.360 (1168.379)
  Night time, Week 12, n=16: number analyzed (Participants) | 16
  Night time, Week 12, n=16 | 280.178 (222.3819)
  Night time, Week 16, n=13: number analyzed (Participants) | 13
  Night time, Week 16, n=13 | 440.992 (641.4221)
  Night time, Week 20, n=13: number analyzed (Participants) | 13
  Night time, Week 20, n=13 | 306.540 (293.6219)
  Night time, Week 24, n=14: number analyzed (Participants) | 14
  Night time, Week 24, n=14 | 442.779 (611.4870)
  Night time, Week 28, n=10: number analyzed (Participants) | 10
  Night time, Week 28, n=10 | 708.219 (967.2115)
  Night time, Week 32, n=12: number analyzed (Participants) | 12
  Night time, Week 32, n=12 | 479.673 (590.4367)
  Night time, Week 36, n=10: number analyzed (Participants) | 10
  Night time, Week 36, n=10 | 462.395 (313.6826)
  Night time, Week 40, n=12: number analyzed (Participants) | 12
  Night time, Week 40, n=12 | 278.703 (264.5554)
  Night time, Week 44, n=11: number analyzed (Participants) | 11
  Night time, Week 44, n=11 | 383.820 (273.3449)
  Night time, Week 48, n=13: number analyzed (Participants) | 13
  Night time, Week 48, n=13 | 493.870 (524.4698)

10. Other Pre Specified Outcome: Mean Maximum Activity Count in a 24 Hour Period
Description: Mean maximum activity count of day time and night time for the 24-hour recording periods; averaged for each time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Count of activity
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Count of activity
  Day time, Week 0, n=24: number analyzed (Participants) | 24
  Day time, Week 0, n=24 | 1618.403 (1288.502)
  Day time, Week 4, n=22: number analyzed (Participants) | 22
  Day time, Week 4, n=22 | 1309.195 (1042.150)
  Day time, Week 8, n=17: number analyzed (Participants) | 17
  Day time, Week 8, n=17 | 1612.785 (1822.405)
  Day time, Week 12, n=16: number analyzed (Participants) | 16
  Day time, Week 12, n=16 | 1165.166 (705.7684)
  Day time, Week 16, n=13: number analyzed (Participants) | 13
  Day time, Week 16, n=13 | 1510.868 (1407.533)
  Day time, Week 20, n=14: number analyzed (Participants) | 14
  Day time, Week 20, n=14 | 1146.578 (1016.899)
  Day time, Week 24, n=13: number analyzed (Participants) | 13
  Day time, Week 24, n=13 | 697.693 (678.2212)
  Day time, Week 28, n=10: number analyzed (Participants) | 10
  Day time, Week 28, n=10 | 665.987 (475.5967)
  Day time, Week 32, n=12: number analyzed (Participants) | 12
  Day time, Week 32, n=12 | 633.595 (536.0698)
  Day time, Week 36, n=12: number analyzed (Participants) | 12
  Day time, Week 36, n=12 | 772.909 (672.3572)
  Day time, Week 40, n=12: number analyzed (Participants) | 12
  Day time, Week 40, n=12 | 543.052 (410.3246)
  Day time, Week 44, n=12: number analyzed (Participants) | 12
  Day time, Week 44, n=12 | 1074.333 (988.7887)
  Day time, Week 48, n=13: number analyzed (Participants) | 13
  Day time, Week 48, n=13 | 1002.060 (1011.468)
  Night time, Week 0, n=24: number analyzed (Participants) | 24
  Night time, Week 0, n=24 | 319.872 (312.3125)
  Night time, Week 4, n=22: number analyzed (Participants) | 22
  Night time, Week 4, n=22 | 231.630 (183.2420)
  Night time, Week 8, n=19: number analyzed (Participants) | 19
  Night time, Week 8, n=19 | 518.646 (1153.825)
  Night time, Week 12, n=16: number analyzed (Participants) | 16
  Night time, Week 12, n=16 | 176.211 (142.6990)
  Night time, Week 16, n=13: number analyzed (Participants) | 13
  Night time, Week 16, n=13 | 194.670 (208.1798)
  Night time, Week 20, n=13: number analyzed (Participants) | 13
  Night time, Week 20, n=13 | 174.990 (153.0679)
  Night time, Week 24, n=14: number analyzed (Participants) | 14
  Night time, Week 24, n=14 | 208.871 (184.5488)
  Night time, Week 28, n=10: number analyzed (Participants) | 10
  Night time, Week 28, n=10 | 325.419 (356.4562)
  Night time, Week 32, n=12: number analyzed (Participants) | 12
  Night time, Week 32, n=12 | 267.311 (294.0265)
  Night time, Week 36, n=10: number analyzed (Participants) | 10
  Night time, Week 36, n=10 | 242.772 (159.5699)
  Night time, Week 40, n=12: number analyzed (Participants) | 12
  Night time, Week 40, n=12 | 145.523 (109.5598)
  Night time, Week 44, n=11: number analyzed (Participants) | 11
  Night time, Week 44, n=11 | 207.506 (134.7506)
  Night time, Week 48, n=13: number analyzed (Participants) | 13
  Night time, Week 48, n=13 | 233.548 (215.7070)

11. Other Pre Specified Outcome: Number of Continuous Active Periods
Description: Active periods were catagorized as >1minute to <=2minutes, >2 minutes to <=5minutes, >5 minutes to <=15 minutes, >15 minutes to <=30 minutes, >30 minutes. Total number of 'active periods were calculated as 1minute<x<2minutes + 'number of active periods 2minutes<x<5minutes + 'number of active periods 5minutes<x<15minutes + 'number of active periods 15minutes<x<30minutes + 'number of active periods >30minutes.
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Number/Hour
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Number/Hour
  >1 to <=2minutes; Day time, Week 0, n=24: number analyzed (Participants) | 24
  >1 to <=2minutes; Day time, Week 0, n=24 | 0.279 (0.3174)
  >1 to <=2minutes;Day time, Week 4, n=22: number analyzed (Participants) | 22
  >1 to <=2minutes;Day time, Week 4, n=22 | 0.267 (0.3874)
  >1 to <=2minutes;Day time, Week 8, n=18: number analyzed (Participants) | 18
  >1 to <=2minutes;Day time, Week 8, n=18 | 0.255 (0.3230)
  >1 to <=2minutes;Day time, Week 12, n=16: number analyzed (Participants) | 16
  >1 to <=2minutes;Day time, Week 12, n=16 | 0.188 (0.1925)
  >1 to <=2minutes;Day time, Week 16, n=13: number analyzed (Participants) | 13
  >1 to <=2minutes;Day time, Week 16, n=13 | 0.191 (0.1996)
  >1 to <=2minutes;Day time, Week 20, n=14: number analyzed (Participants) | 14
  >1 to <=2minutes;Day time, Week 20, n=14 | 0.169 (0.1812)
  >1 to <=2minutes;Day time, Week 24, n=14: number analyzed (Participants) | 14
  >1 to <=2minutes;Day time, Week 24, n=14 | 0.206 (0.2088)
  >1 to <=2minutes;Day time, Week 28, n=10: number analyzed (Participants) | 10
  >1 to <=2minutes;Day time, Week 28, n=10 | 0.147 (0.1564)
  >1 to <=2minutes;Day time, Week 32, n=12: number analyzed (Participants) | 12
  >1 to <=2minutes;Day time, Week 32, n=12 | 0.100 (0.1172)
  >1 to <=2minutes;Day time, Week 36, n=12: number analyzed (Participants) | 12
  >1 to <=2minutes;Day time, Week 36, n=12 | 0.164 (0.2649)
  >1 to <=2minutes;Day time, Week 40, n=12: number analyzed (Participants) | 12
  >1 to <=2minutes;Day time, Week 40, n=12 | 0.170 (0.2644)
  >1 to <=2minutes;Day time, Week 44, n=12: number analyzed (Participants) | 12
  >1 to <=2minutes;Day time, Week 44, n=12 | 0.174 (0.2518)
  >1 to <=2minutes;Day time, Week 48, n=13: number analyzed (Participants) | 13
  >1 to <=2minutes;Day time, Week 48, n=13 | 0.252 (0.3609)
  >2 to <=5minutes; Day time, Week 0, n=24: number analyzed (Participants) | 24
  >2 to <=5minutes; Day time, Week 0, n=24 | 0.108 (0.1263)
  >2 to <=5minutes;Day time, Week 4, n=22: number analyzed (Participants) | 22
  >2 to <=5minutes;Day time, Week 4, n=22 | 0.097 (0.1264)
  >2 to <=5minutes;Day time, Week 8, n=18: number analyzed (Participants) | 18
  >2 to <=5minutes;Day time, Week 8, n=18 | 0.084 (0.1675)
  >2 to <=5minutes;Day time, Week 12, n=16: number analyzed (Participants) | 16
  >2 to <=5minutes;Day time, Week 12, n=16 | 0.108 (0.1201)
  >2 to <=5minutes;Day time, Week 16, n=13: number analyzed (Participants) | 13
  >2 to <=5minutes;Day time, Week 16, n=13 | 0.123 (0.1590)
  >2 to <=5minutes;Day time, Week 20, n=14: number analyzed (Participants) | 14
  >2 to <=5minutes;Day time, Week 20, n=14 | 0.080 (0.1105)
  >2 to <=5minutes;Day time, Week 24, n=14: number analyzed (Participants) | 14
  >2 to <=5minutes;Day time, Week 24, n=14 | 0.057 (0.0819)
  >2 to <=5minutes;Day time, Week 28, n=10: number analyzed (Participants) | 10
  >2 to <=5minutes;Day time, Week 28, n=10 | 0.107 (0.1700)
  >2 to <=5minutes;Day time, Week 32, n=12: number analyzed (Participants) | 12
  >2 to <=5minutes;Day time, Week 32, n=12 | 0.058 (0.1129)
  >2 to <=5minutes;Day time, Week 36, n=12: number analyzed (Participants) | 12
  >2 to <=5minutes;Day time, Week 36, n=12 | 0.079 (0.1538)
  >2 to <=5minutes;Day time, Week 40, n=12: number analyzed (Participants) | 12
  >2 to <=5minutes;Day time, Week 40, n=12 | 0.072 (0.1137)
  >2 to <=5minutes;Day time, Week 44, n=12: number analyzed (Participants) | 12
  >2 to <=5minutes;Day time, Week 44, n=12 | 0.071 (0.1417)
  >2 to <=5minutes;Day time, Week 48, n=13: number analyzed (Participants) | 13
  >2 to <=5minutes;Day time, Week 48, n=13 | 0.095 (0.1400)
  >5 to <=15 minutes; Day time, Week 0, n=24: number analyzed (Participants) | 24
  >5 to <=15 minutes; Day time, Week 0, n=24 | 0.041 (0.0740)
  >5 to <=15 minutes;Day time, Week 4, n=22: number analyzed (Participants) | 22
  >5 to <=15 minutes;Day time, Week 4, n=22 | 0.030 (0.0471)
  >5 to <=15 minutes;Day time, Week 8, n=18: number analyzed (Participants) | 18
  >5 to <=15 minutes;Day time, Week 8, n=18 | 0.020 (0.0333)
  >5 to <=15 minutes;Day time, Week 12, n=16: number analyzed (Participants) | 16
  >5 to <=15 minutes;Day time, Week 12, n=16 | 0.023 (0.0364)
  >5 to <=15 minutes;Day time, Week 16, n=13: number analyzed (Participants) | 13
  >5 to <=15 minutes;Day time, Week 16, n=13 | 0.042 (0.0699)
  >5 to <=15 minutes;Day time, Week 20, n=14: number analyzed (Participants) | 14
  >5 to <=15 minutes;Day time, Week 20, n=14 | 0.016 (0.0440)
  >5 to <=15 minutes;Day time, Week 24, n=14: number analyzed (Participants) | 14
  >5 to <=15 minutes;Day time, Week 24, n=14 | 0.000 (0.000)
  >5 to <=15 minutes;Day time, Week 28, n=10: number analyzed (Participants) | 10
  >5 to <=15 minutes;Day time, Week 28, n=10 | 0.024 (0.0534)
  >5 to <=15 minutes;Day time, Week 32, n=12: number analyzed (Participants) | 12
  >5 to <=15 minutes;Day time, Week 32, n=12 | 0.015 (0.0353)
  >5 to <=15 minutes;Day time, Week 36, n=12: number analyzed (Participants) | 12
  >5 to <=15 minutes;Day time, Week 36, n=12 | 0.008 (0.0289)
  >5 to <=15 minutes;Day time, Week 40, n=12: number analyzed (Participants) | 12
  >5 to <=15 minutes;Day time, Week 40, n=12 | 0.022 (0.0549)
  >5 to <=15 minutes;Day time, Week 44, n=12: number analyzed (Participants) | 12
  >5 to <=15 minutes;Day time, Week 44, n=12 | 0.008 (0.0199)
  >5 to <=15 minutes;Day time, Week 48, n=13: number analyzed (Participants) | 13
  >5 to <=15 minutes;Day time, Week 48, n=13 | 0.023 (0.0440)
  >15 to <=30 minutes; Day time, Week 0, n=24: number analyzed (Participants) | 24
  >15 to <=30 minutes; Day time, Week 0, n=24 | 0.003 (0.0108)
  >15 to <=30 minutes;Day time, Week 4, n=22: number analyzed (Participants) | 22
  >15 to <=30 minutes;Day time, Week 4, n=22 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 8, n=18: number analyzed (Participants) | 18
  >15 to <=30 minutes;Day time, Week 8, n=18 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 12, n=16: number analyzed (Participants) | 16
  >15 to <=30 minutes;Day time, Week 12, n=16 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 16, n=13: number analyzed (Participants) | 13
  >15 to <=30 minutes;Day time, Week 16, n=13 | 0.003 (0.0111)
  >15 to <=30 minutes;Day time, Week 20, n=14: number analyzed (Participants) | 14
  >15 to <=30 minutes;Day time, Week 20, n=14 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 24, n=14: number analyzed (Participants) | 14
  >15 to <=30 minutes;Day time, Week 24, n=14 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 28, n=10: number analyzed (Participants) | 10
  >15 to <=30 minutes;Day time, Week 28, n=10 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 32, n=12: number analyzed (Participants) | 12
  >15 to <=30 minutes;Day time, Week 32, n=12 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 36, n=12: number analyzed (Participants) | 12
  >15 to <=30 minutes;Day time, Week 36, n=12 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 40, n=12: number analyzed (Participants) | 12
  >15 to <=30 minutes;Day time, Week 40, n=12 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 44, n=12: number analyzed (Participants) | 12
  >15 to <=30 minutes;Day time, Week 44, n=12 | 0.000 (0.000)
  >15 to <=30 minutes;Day time, Week 48, n=13: number analyzed (Participants) | 13
  >15 to <=30 minutes;Day time, Week 48, n=13 | 0.000 (0.000)
  >30 minutes; Day time, Week 0, n=24: number analyzed (Participants) | 24
  >30 minutes; Day time, Week 0, n=24 | 0.000 (0.000)
  >30 minutes;Day time, Week 4, n=22: number analyzed (Participants) | 22
  >30 minutes;Day time, Week 4, n=22 | 0.000 (0.000)
  >30 minutes;Day time, Week 8, n=18: number analyzed (Participants) | 18
  >30 minutes;Day time, Week 8, n=18 | 0.001 (0.0047)
  >30 minutes;Day time, Week 12, n=16: number analyzed (Participants) | 16
  >30 minutes;Day time, Week 12, n=16 | 0.000 (0.000)
  >30 minutes;Day time, Week 16, n=13: number analyzed (Participants) | 13
  >30 minutes;Day time, Week 16, n=13 | 0.000 (0.000)
  >30 minutes;Day time, Week 20, n=14: number analyzed (Participants) | 14
  >30 minutes;Day time, Week 20, n=14 | 0.000 (0.000)
  >30 minutes;Day time, Week 24, n=14: number analyzed (Participants) | 14
  >30 minutes;Day time, Week 24, n=14 | 0.000 (0.000)
  >30 minutes;Day time, Week 28, n=10: number analyzed (Participants) | 10
  >30 minutes;Day time, Week 28, n=10 | 0.000 (0.000)
  >30 minutes;Day time, Week 32, n=12: number analyzed (Participants) | 12
  >30 minutes;Day time, Week 32, n=12 | 0.000 (0.000)
  >30 minutes;Day time, Week 36, n=12: number analyzed (Participants) | 12
  >30 minutes;Day time, Week 36, n=12 | 0.000 (0.000)
  >30 minutes;Day time, Week 40, n=12: number analyzed (Participants) | 12
  >30 minutes;Day time, Week 40, n=12 | 0.000 (0.000)
  >30 minutes;Day time, Week 44, n=12: number analyzed (Participants) | 12
  >30 minutes;Day time, Week 44, n=12 | 0.000 (0.000)
  >30 minutes;Day time, Week 48, n=13: number analyzed (Participants) | 13
  >30 minutes;Day time, Week 48, n=13 | 0.000 (0.000)
  >1 to <=2minutes; Night time, Week 0, n=24: number analyzed (Participants) | 24
  >1 to <=2minutes; Night time, Week 0, n=24 | 0.015 (0.0365)
  >1 to <=2minutes;Night time, Week 4, n=22: number analyzed (Participants) | 22
  >1 to <=2minutes;Night time, Week 4, n=22 | 0.000 (0.000)
  >1 to <=2minutes;Night time, Week 8, n=19: number analyzed (Participants) | 19
  >1 to <=2minutes;Night time, Week 8, n=19 | 0.046 (0.1453)
  >1 to <=2minutes;Night time, Week 12, n=16: number analyzed (Participants) | 16
  >1 to <=2minutes;Night time, Week 12, n=16 | 0.000 (0.000)
  >1 to <=2minutes;Night time, Week 16, n=13: number analyzed (Participants) | 13
  >1 to <=2minutes;Night time, Week 16, n=13 | 0.000 (0.000)
  >1 to <=2minutes;Night time, Week 20, n=13: number analyzed (Participants) | 13
  >1 to <=2minutes;Night time, Week 20, n=13 | 0.003 (0.0111)
  >1 to <=2minutes;Night time, Week 24, n=14: number analyzed (Participants) | 14
  >1 to <=2minutes;Night time, Week 24, n=14 | 0.000 (0.000)
  >1 to <=2minutes;Night time, Week 28, n=10: number analyzed (Participants) | 10
  >1 to <=2minutes;Night time, Week 28, n=10 | 0.004 (0.0126)
  >1 to <=2minutes;Night time, Week 32, n=12: number analyzed (Participants) | 12
  >1 to <=2minutes;Night time, Week 32, n=12 | 0.004 (0.0144)
  >1 to <=2minutes;Night time, Week 36, n=10: number analyzed (Participants) | 10
  >1 to <=2minutes;Night time, Week 36, n=10 | 0.000 (0.000)
  >1 to <=2minutes;Night time, Week 40, n=12: number analyzed (Participants) | 12
  >1 to <=2minutes;Night time, Week 40, n=12 | 0.000 (0.000)
  >1 to <=2minutes;Night time, Week 44, n=11: number analyzed (Participants) | 11
  >1 to <=2minutes;Night time, Week 44, n=11 | 0.000 (0.000)
  >1 to <=2minutes;Night time, Week 48, n=13: number analyzed (Participants) | 13
  >1 to <=2minutes;Night time, Week 48, n=13 | 0.292 (1.0512)
  >2 to <=5minutes; Night time, Week 0, n=24: number analyzed (Participants) | 24
  >2 to <=5minutes; Night time, Week 0, n=24 | 0.008 (0.0284)
  >2 to <=5minutes;Night time, Week 4, n=22: number analyzed (Participants) | 22
  >2 to <=5minutes;Night time, Week 4, n=22 | 0.000 (0.000)
  >2 to <=5minutes;Night time, Week 8, n=19: number analyzed (Participants) | 19
  >2 to <=5minutes;Night time, Week 8, n=19 | 0.067 (0.2617)
  >2 to <=5minutes;Night time, Week 12, n=16: number analyzed (Participants) | 16
  >2 to <=5minutes;Night time, Week 12, n=16 | 0.000 (0.000)
  >2 to <=5minutes;Night time, Week 16, n=13: number analyzed (Participants) | 13
  >2 to <=5minutes;Night time, Week 16, n=13 | 0.000 (0.000)
  >2 to <=5minutes;Night time, Week 20, n=13: number analyzed (Participants) | 13
  >2 to <=5minutes;Night time, Week 20, n=13 | 0.000 (0.000)
  >2 to <=5minutes;Night time, Week 24, n=14: number analyzed (Participants) | 14
  >2 to <=5minutes;Night time, Week 24, n=14 | 0.000 (0.000)
  >2 to <=5minutes;Night time, Week 28, n=10: number analyzed (Participants) | 10
  >2 to <=5minutes;Night time, Week 28, n=10 | 0.006 (0.0190)
  >2 to <=5minutes;Night time, Week 32, n=12: number analyzed (Participants) | 12
  >2 to <=5minutes;Night time, Week 32, n=12 | 0.000 (0.000)
  >2 to <=5minutes;Night time, Week 36, n=10: number analyzed (Participants) | 10
  >2 to <=5minutes;Night time, Week 36, n=10 | 0.000 (0.000)
  >2 to <=5minutes;Night time, Week 40, n=12: number analyzed (Participants) | 12
  >2 to <=5minutes;Night time, Week 40, n=12 | 0.000 (0.000)
  >2 to <=5minutes;Night time, Week 44, n=11: number analyzed (Participants) | 11
  >2 to <=5minutes;Night time, Week 44, n=11 | 0.000 (0.000)
  >2 to <=5minutes;Night time, Week 48, n=13: number analyzed (Participants) | 13
  >2 to <=5minutes;Night time, Week 48, n=13 | 0.000 (0.000)
  >5 to <=15 minutes; Night time, Week 0, n=24: number analyzed (Participants) | 24
  >5 to <=15 minutes; Night time, Week 0, n=24 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 4, n=22: number analyzed (Participants) | 22
  >5 to <=15 minutes;Night time, Week 4, n=22 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 8, n=19: number analyzed (Participants) | 19
  >5 to <=15 minutes;Night time, Week 8, n=19 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 12, n=16: number analyzed (Participants) | 16
  >5 to <=15 minutes;Night time, Week 12, n=16 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 16, n=13: number analyzed (Participants) | 13
  >5 to <=15 minutes;Night time, Week 16, n=13 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 20, n=13: number analyzed (Participants) | 13
  >5 to <=15 minutes;Night time, Week 20, n=13 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 24, n=14: number analyzed (Participants) | 14
  >5 to <=15 minutes;Night time, Week 24, n=14 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 28, n=10: number analyzed (Participants) | 10
  >5 to <=15 minutes;Night time, Week 28, n=10 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 32, n=12: number analyzed (Participants) | 12
  >5 to <=15 minutes;Night time, Week 32, n=12 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 36, n=10: number analyzed (Participants) | 10
  >5 to <=15 minutes;Night time, Week 36, n=10 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 40, n=12: number analyzed (Participants) | 12
  >5 to <=15 minutes;Night time, Week 40, n=12 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 44, n=11: number analyzed (Participants) | 11
  >5 to <=15 minutes;Night time, Week 44, n=11 | 0.000 (0.000)
  >5 to <=15 minutes;Night time, Week 48, n=13: number analyzed (Participants) | 13
  >5 to <=15 minutes;Night time, Week 48, n=13 | 0.000 (0.000)
  >15 to <=30 minutes; Night time, Week 0, n=24: number analyzed (Participants) | 24
  >15 to <=30 minutes; Night time, Week 0, n=24 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 4, n=22: number analyzed (Participants) | 22
  >15 to <=30 minutes;Night time, Week 4, n=22 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 8, n=19: number analyzed (Participants) | 19
  >15 to <=30 minutes;Night time, Week 8, n=19 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 12, n=16: number analyzed (Participants) | 16
  >15 to <=30 minutes;Night time, Week 12, n=16 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 16, n=13: number analyzed (Participants) | 13
  >15 to <=30 minutes;Night time, Week 16, n=13 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 20, n=13: number analyzed (Participants) | 13
  >15 to <=30 minutes;Night time, Week 20, n=13 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 24, n=14: number analyzed (Participants) | 14
  >15 to <=30 minutes;Night time, Week 24, n=14 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 28, n=10: number analyzed (Participants) | 10
  >15 to <=30 minutes;Night time, Week 28, n=10 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 32, n=12: number analyzed (Participants) | 12
  >15 to <=30 minutes;Night time, Week 32, n=12 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 36, n=10: number analyzed (Participants) | 10
  >15 to <=30 minutes;Night time, Week 36, n=10 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 40, n=12: number analyzed (Participants) | 12
  >15 to <=30 minutes;Night time, Week 40, n=12 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 44, n=11: number analyzed (Participants) | 11
  >15 to <=30 minutes;Night time, Week 44, n=11 | 0.000 (0.000)
  >15 to <=30 minutes;Night time, Week 48, n=13: number analyzed (Participants) | 13
  >15 to <=30 minutes;Night time, Week 48, n=13 | 0.000 (0.000)
  >30 minutes; Night time, Week 0, n=24: number analyzed (Participants) | 24
  >30 minutes; Night time, Week 0, n=24 | 0.000 (0.000)
  >30 minutes;Night time, Week 4, n=22: number analyzed (Participants) | 22
  >30 minutes;Night time, Week 4, n=22 | 0.000 (0.000)
  >30 minutes;Night time, Week 8, n=19: number analyzed (Participants) | 19
  >30 minutes;Night time, Week 8, n=19 | 0.000 (0.000)
  >30 minutes;Night time, Week 12, n=16: number analyzed (Participants) | 16
  >30 minutes;Night time, Week 12, n=16 | 0.000 (0.000)
  >30 minutes;Night time, Week 16, n=13: number analyzed (Participants) | 13
  >30 minutes;Night time, Week 16, n=13 | 0.000 (0.000)
  >30 minutes;Night time, Week 20, n=13: number analyzed (Participants) | 13
  >30 minutes;Night time, Week 20, n=13 | 0.000 (0.000)
  >30 minutes;Night time, Week 24, n=14: number analyzed (Participants) | 14
  >30 minutes;Night time, Week 24, n=14 | 0.000 (0.000)
  >30 minutes;Night time, Week 28, n=10: number analyzed (Participants) | 10
  >30 minutes;Night time, Week 28, n=10 | 0.000 (0.000)
  >30 minutes;Night time, Week 32, n=12: number analyzed (Participants) | 12
  >30 minutes;Night time, Week 32, n=12 | 0.000 (0.000)
  >30 minutes;Night time, Week 36, n=10: number analyzed (Participants) | 10
  >30 minutes;Night time, Week 36, n=10 | 0.000 (0.000)
  >30 minutes;Night time, Week 40, n=12: number analyzed (Participants) | 12
  >30 minutes;Night time, Week 40, n=12 | 0.000 (0.000)
  >30 minutes;Night time, Week 44, n=11: number analyzed (Participants) | 11
  >30 minutes;Night time, Week 44, n=11 | 0.000 (0.000)
  >30 minutes;Night time, Week 48, n=13: number analyzed (Participants) | 13
  >30 minutes;Night time, Week 48, n=13 | 0.000 (0.000)

12. Other Pre Specified Outcome: Percent of Time Lying Down at Night
Description: Percent time spent lying per day and night over the 24-hour recording periods; averaged for each timepoint
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Percentage of time
  Day time, Week 0, n=24: number analyzed (Participants) | 24
  Day time, Week 0, n=24 | 12.079 (8.3771)
  Day time, Week 4, n=22: number analyzed (Participants) | 22
  Day time, Week 4, n=22 | 14.119 (13.8340)
  Day time, Week 8, n=18: number analyzed (Participants) | 18
  Day time, Week 8, n=18 | 17.993 (12.7684)
  Day time, Week 12, n=16: number analyzed (Participants) | 16
  Day time, Week 12, n=16 | 13.101 (9.7891)
  Day time, Week 16, n=13: number analyzed (Participants) | 13
  Day time, Week 16, n=13 | 12.400 (9.3903)
  Day time, Week 20, n=14: number analyzed (Participants) | 14
  Day time, Week 20, n=14 | 21.198 (25.9982)
  Day time, Week 24, n=14: number analyzed (Participants) | 14
  Day time, Week 24, n=14 | 23.608 (28.1925)
  Day time, Week 28, n=10: number analyzed (Participants) | 10
  Day time, Week 28, n=10 | 23.603 (23.9283)
  Day time, Week 32, n=12: number analyzed (Participants) | 12
  Day time, Week 32, n=12 | 26.613 (34.2248)
  Day time, Week 36, n=12: number analyzed (Participants) | 12
  Day time, Week 36, n=12 | 21.823 (28.2251)
  Day time, Week 40, n=12: number analyzed (Participants) | 12
  Day time, Week 40, n=12 | 17.453 (19.6178)
  Day time, Week 44, n=12: number analyzed (Participants) | 12
  Day time, Week 44, n=12 | 20.397 (26.7615)
  Day time, Week 48, n=13: number analyzed (Participants) | 13
  Day time, Week 48, n=13 | 20.966 (20.3006)
  Night time, Week 0, n=24: number analyzed (Participants) | 24
  Night time, Week 0, n=24 | 95.131 (8.2933)
  Night time, Week 4, n=22: number analyzed (Participants) | 22
  Night time, Week 4, n=22 | 97.280 (2.9257)
  Night time, Week 8, n=19: number analyzed (Participants) | 19
  Night time, Week 8, n=19 | 96.871 (4.0262)
  Night time, Week 12, n=16: number analyzed (Participants) | 16
  Night time, Week 12, n=16 | 97.886 (1.4457)
  Night time, Week 16, n=13: number analyzed (Participants) | 13
  Night time, Week 16, n=13 | 97.817 (1.1466)
  Night time, Week 20, n=13: number analyzed (Participants) | 13
  Night time, Week 20, n=13 | 97.739 (1.1617)
  Night time, Week 24, n=14: number analyzed (Participants) | 14
  Night time, Week 24, n=14 | 97.522 (1.6446)
  Night time, Week 28, n=10: number analyzed (Participants) | 10
  Night time, Week 28, n=10 | 96.397 (2.1777)
  Night time, Week 32, n=12: number analyzed (Participants) | 12
  Night time, Week 32, n=12 | 95.519 (6.0885)
  Night time, Week 36, n=10: number analyzed (Participants) | 10
  Night time, Week 36, n=10 | 98.165 (0.6796)
  Night time, Week 40, n=12: number analyzed (Participants) | 12
  Night time, Week 40, n=12 | 97.293 (1.8971)
  Night time, Week 44, n=11: number analyzed (Participants) | 11
  Night time, Week 44, n=11 | 97.719 (1.6543)
  Night time, Week 48, n=13: number analyzed (Participants) | 13
  Night time, Week 48, n=13 | 93.912 (14.0863)

13. Other Pre Specified Outcome: Number of Night Time Movement Episodes Per Hour
Description: Average number of night movement episodes per hour for each protocol time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Number of movements/hour
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Number of movements/hour
  Week 0, n=24: number analyzed (Participants) | 24
  Week 0, n=24 | 6.129 (4.6585)
  Week 4, n=22: number analyzed (Participants) | 22
  Week 4, n=22 | 6.982 (7.6835)
  Week 8, n=19: number analyzed (Participants) | 19
  Week 8, n=19 | 9.258 (17.3296)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 3.803 (1.7339)
  Week 16, n=13: number analyzed (Participants) | 13
  Week 16, n=13 | 6.852 (11.6765)
  Week 20, n=13: number analyzed (Participants) | 13
  Week 20, n=13 | 4.788 (4.4738)
  Week 24, n=14: number analyzed (Participants) | 14
  Week 24, n=14 | 4.216 (1.8617)
  Week 28, n=10: number analyzed (Participants) | 10
  Week 28, n=10 | 5.295 (5.1177)
  Week 32, n=12: number analyzed (Participants) | 12
  Week 32, n=12 | 8.708 (12.9217)
  Week 36, n=10: number analyzed (Participants) | 10
  Week 36, n=10 | 12.149 (17.7170)
  Week 40, n=12: number analyzed (Participants) | 12
  Week 40, n=12 | 4.747 (4.5737)
  Week 44, n=11: number analyzed (Participants) | 11
  Week 44, n=11 | 3.385 (1.8031)
  Week 48, n=13: number analyzed (Participants) | 13
  Week 48, n=13 | 7.209 (13.6287)

14. Other Pre Specified Outcome: Percent Time Night-time Rest Efficiency
Description: Average night-time rest efficiency for each protocol time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Percentage of time
  Week 0, n=24: number analyzed (Participants) | 24
  Week 0, n=24 | 0.986 (0.0125)
  Week 4, n=22: number analyzed (Participants) | 22
  Week 4, n=22 | 0.982 (0.0270)
  Week 8, n=19: number analyzed (Participants) | 19
  Week 8, n=19 | 0.976 (0.0498)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 0.991 (0.0044)
  Week 16, n=13: number analyzed (Participants) | 13
  Week 16, n=13 | 0.986 (0.0156)
  Week 20, n=13: number analyzed (Participants) | 13
  Week 20, n=13 | 0.987 (0.0118)
  Week 24, n=14: number analyzed (Participants) | 14
  Week 24, n=14 | 0.991 (0.0053)
  Week 28, n=10: number analyzed (Participants) | 10
  Week 28, n=10 | 0.986 (0.0165)
  Week 32, n=12: number analyzed (Participants) | 12
  Week 32, n=12 | 0.978 (0.0322)
  Week 36, n=10: number analyzed (Participants) | 10
  Week 36, n=10 | 0.971 (0.0468)
  Week 40, n=12: number analyzed (Participants) | 12
  Week 40, n=12 | 0.987 (0.0156)
  Week 44, n=11: number analyzed (Participants) | 11
  Week 44, n=11 | 0.992 (0.0040)
  Week 48, n=13: number analyzed (Participants) | 13
  Week 48, n=13 | 0.978 (0.0536)

15. Other Pre Specified Outcome: Rest Fragmentation Index
Description: Rest Fragmentation Index was computed as movement time (%) divided by number of movement episodes for each protocol time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0, n=24: number analyzed (Participants) | 24
  Week 0, n=24 | 0.132 (0.3384)
  Week 4, n=22: number analyzed (Participants) | 22
  Week 4, n=22 | 0.649 (2.6064)
  Week 8, n=19: number analyzed (Participants) | 19
  Week 8, n=19 | 0.096 (0.2579)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 0.036 (0.0316)
  Week 16, n=13: number analyzed (Participants) | 13
  Week 16, n=13 | 0.291 (0.8315)
  Week 20, n=13: number analyzed (Participants) | 13
  Week 20, n=13 | 0.086 (0.1581)
  Week 24, n=14: number analyzed (Participants) | 14
  Week 24, n=14 | 0.129 (0.3213)
  Week 28, n=10: number analyzed (Participants) | 10
  Week 28, n=10 | 0.113 (0.2836)
  Week 32, n=12: number analyzed (Participants) | 12
  Week 32, n=12 | 0.507 (1.1908)
  Week 36, n=10: number analyzed (Participants) | 10
  Week 36, n=10 | 0.437 (1.1594)
  Week 40, n=12: number analyzed (Participants) | 12
  Week 40, n=12 | 0.541 (1.7070)
  Week 44, n=11: number analyzed (Participants) | 11
  Week 44, n=11 | 0.041 (0.0259)
  Week 48, n=13: number analyzed (Participants) | 13
  Week 48, n=13 | 0.391 (1.2979)

16. Other Pre Specified Outcome: Average Duration of Night Time Movement Episodes
Description: Average duration of movement episodes for each time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Seconds
  Week 0, n=24: number analyzed (Participants) | 24
  Week 0, n=24 | 8.257 (2.5147)
  Week 4, n=22: number analyzed (Participants) | 22
  Week 4, n=22 | 7.664 (2.0949)
  Week 8, n=19: number analyzed (Participants) | 19
  Week 8, n=19 | 8.133 (2.8630)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 8.203 (2.3391)
  Week 16, n=13: number analyzed (Participants) | 13
  Week 16, n=13 | 9.485 (5.4216)
  Week 20, n=13: number analyzed (Participants) | 13
  Week 20, n=13 | 10.190 (7.2948)
  Week 24, n=14: number analyzed (Participants) | 14
  Week 24, n=14 | 7.931 (1.8877)
  Week 28, n=10: number analyzed (Participants) | 10
  Week 28, n=10 | 7.610 (1.5252)
  Week 32, n=11: number analyzed (Participants) | 11
  Week 32, n=11 | 10.220 (6.3726)
  Week 36, n=9: number analyzed (Participants) | 9
  Week 36, n=9 | 7.203 (0.6451)
  Week 40, n=11: number analyzed (Participants) | 11
  Week 40, n=11 | 8.025 (1.8174)
  Week 44, n=11: number analyzed (Participants) | 11
  Week 44, n=11 | 7.730 (2.3985)
  Week 48, n=12: number analyzed (Participants) | 12
  Week 48, n=12 | 8.393 (2.5605)

17. Other Pre Specified Outcome: Relationship Between Average Number Night Time Movements/Hour Versus Total ALSFRS-R
Description: Estimates for between and within subject correlation coefficients were produced following multiple linear regression analyses on the actigraphy endpoints, comparing them with the ALSFRS-R total score and the gross motor domain and fine motor domain scores. Data for between subject correlation coefficient has been presented
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio | 0.178

18. Other Pre Specified Outcome: Relationship Between Average Duration Movement Episodes at Night Versus Total ALSFRS-R
Description: as for outcome 17
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio | -0.426

19. Other Pre Specified Outcome: Relationship Between Average Percent Time Night Time Rest Efficiency Versus Total ALSFRS-R
Description: as for outcome 17
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio | 0.049

20. Other Pre Specified Outcome: Relationship Between Average Night Time Rest Fragmentation Index Versus Total ALSFRS-R
Description: as for outcome 17
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio | -0.163

21. Other Pre Specified Outcome: Mean Heart Rate Variability (HRV) While Lying (Low Frequency[LF]/High Frequency[HF])
Description: Mean Heart Rate Variability (HRV) averaged over 5 windows of lying down at each protocol time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0, n=23: number analyzed (Participants) | 23
  Week 0, n=23 | 4.1914 (2.35370)
  Week 4, n=21: number analyzed (Participants) | 21
  Week 4, n=21 | 4.2198 (2.88326)
  Week 8, n=15: number analyzed (Participants) | 15
  Week 8, n=15 | 4.2393 (2.50840)
  Week 12, n=15: number analyzed (Participants) | 15
  Week 12, n=15 | 4.2304 (2.13905)
  Week 16, n=12: number analyzed (Participants) | 12
  Week 16, n=12 | 3.7404 (1.99810)
  Week 20, n=12: number analyzed (Participants) | 12
  Week 20, n=12 | 4.6210 (3.40720)
  Week 24, n=12: number analyzed (Participants) | 12
  Week 24, n=12 | 4.2944 (2.43365)
  Week 28, n=10: number analyzed (Participants) | 10
  Week 28, n=10 | 6.1888 (5.64815)
  Week 32, n=10: number analyzed (Participants) | 10
  Week 32, n=10 | 5.0398 (3.64394)
  Week 36, n=9: number analyzed (Participants) | 9
  Week 36, n=9 | 4.9206 (3.44514)
  Week 40, n=11: number analyzed (Participants) | 11
  Week 40, n=11 | 4.6117 (2.81758)
  Week 44, n=11: number analyzed (Participants) | 11
  Week 44, n=11 | 3.8315 (2.29689)
  Week 48, n=11: number analyzed (Participants) | 11
  Week 48, n=11 | 4.4358 (2.56115)

22. Other Pre Specified Outcome: Variance of HRV While Lying (LF/HF)
Description: Variance of Heart Rate Variability (HRV) averaged over 5 windows of lying down at each protocol time point (LF/HF analysis). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0, n=23: number analyzed (Participants) | 23
  Week 0, n=23 | 6.3439 (6.55782)
  Week 4, n=21: number analyzed (Participants) | 21
  Week 4, n=21 | 6.8401 (6.49766)
  Week 8, n=15: number analyzed (Participants) | 15
  Week 8, n=15 | 5.3481 (4.86394)
  Week 12, n=15: number analyzed (Participants) | 15
  Week 12, n=15 | 11.4190 (11.42238)
  Week 16, n=12: number analyzed (Participants) | 12
  Week 16, n=12 | 16.1974 (20.59606)
  Week 20, n=12: number analyzed (Participants) | 12
  Week 20, n=12 | 10.2248 (13.69276)
  Week 24, n=12: number analyzed (Participants) | 12
  Week 24, n=12 | 6.5774 (9.07676)
  Week 28, n=10: number analyzed (Participants) | 10
  Week 28, n=10 | 6.6424 (7.53794)
  Week 32, n=10: number analyzed (Participants) | 10
  Week 32, n=10 | 5.8556 (7.19624)
  Week 36, n=9: number analyzed (Participants) | 9
  Week 36, n=9 | 15.4940 (30.00587)
  Week 40, n=11: number analyzed (Participants) | 11
  Week 40, n=11 | 4.5088 (3.56720)
  Week 44, n=11: number analyzed (Participants) | 11
  Week 44, n=11 | 6.4731 (6.29614)
  Week 48, n=11: number analyzed (Participants) | 11
  Week 48, n=11 | 11.7375 (13.64105)

23. Other Pre Specified Outcome: Mean HRV While Sedentary Not Lying (LF/HF)
Description: Mean Heart Rate Variability (HRV) averaged over 5 windows of sedentary not lying at each protocol time point (LF/HF analysis). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0, n=20: number analyzed (Participants) | 20
  Week 0, n=20 | 5.2011 (2.48369)
  Week 4, n=18: number analyzed (Participants) | 18
  Week 4, n=18 | 5.3944 (2.83547)
  Week 8, n=13: number analyzed (Participants) | 13
  Week 8, n=13 | 5.1733 (2.29737)
  Week 12, n=14: number analyzed (Participants) | 14
  Week 12, n=14 | 6.3760 (3.42063)
  Week 16, n=11: number analyzed (Participants) | 11
  Week 16, n=11 | 6.0905 (3.68543)
  Week 20, n=10: number analyzed (Participants) | 10
  Week 20, n=10 | 6.0958 (3.05182)
  Week 24, n=10: number analyzed (Participants) | 10
  Week 24, n=10 | 6.3113 (3.03599)
  Week 28, n=9: number analyzed (Participants) | 9
  Week 28, n=9 | 5.4652 (3.20703)
  Week 32, n=9: number analyzed (Participants) | 9
  Week 32, n=9 | 8.3196 (5.37661)
  Week 36, n=11: number analyzed (Participants) | 11
  Week 36, n=11 | 6.6827 (2.73499)
  Week 40, n=9: number analyzed (Participants) | 9
  Week 40, n=9 | 4.8166 (2.16486)
  Week 44, n=9: number analyzed (Participants) | 9
  Week 44, n=9 | 5.6220 (2.61752)
  Week 48, n=7: number analyzed (Participants) | 7
  Week 48, n=7 | 5.8935 (3.22033)

24. Other Pre Specified Outcome: Variance of HRV While Sedentary Not Lying (LF/HF)
Description: Variance of Heart Rate Variability (HRV) averaged over 5 windows of sedentary not lying at each protocol time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0, n=20: number analyzed (Participants) | 20
  Week 0, n=20 | 6.3439 (6.55782)
  Week 4, n=18: number analyzed (Participants) | 18
  Week 4, n=18 | 6.8401 (6.49766)
  Week 8, n=13: number analyzed (Participants) | 13
  Week 8, n=13 | 5.3481 (4.86394)
  Week 12, n=14: number analyzed (Participants) | 14
  Week 12, n=14 | 11.4190 (11.42238)
  Week 16, n=11: number analyzed (Participants) | 11
  Week 16, n=11 | 16.1974 (20.59606)
  Week 20, n=10: number analyzed (Participants) | 10
  Week 20, n=10 | 10.2248 (13.69276)
  Week 24, n=10: number analyzed (Participants) | 10
  Week 24, n=10 | 6.5774 (9.07676)
  Week 28, n=9: number analyzed (Participants) | 9
  Week 28, n=9 | 6.6424 (7.53794)
  Week 32, n=9: number analyzed (Participants) | 9
  Week 32, n=9 | 5.8556 (7.19624)
  Week 36, n=11: number analyzed (Participants) | 11
  Week 36, n=11 | 15.4940 (30.00587)
  Week 40, n=9: number analyzed (Participants) | 9
  Week 40, n=9 | 4.5088 (3.56720)
  Week 44, n=9: number analyzed (Participants) | 9
  Week 44, n=9 | 6.4731 (6.29614)
  Week 48, n=7: number analyzed (Participants) | 7
  Week 48, n=7 | 11.7375 (13.64105)

25. Other Pre Specified Outcome: Mean HRV While Active (LF/HF)
Description: Mean Heart Rate Variability (HRV) averaged over 5 windows of subjects being active at each protocol time point (LF/HF analysis). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data is not available. Standard deviation could not be calculated when number of participants was <=1
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0, n=2: number analyzed (Participants) | 2
  Week 0, n=2 | 4.3350 (0.09192)
  Week 4, n=1: number analyzed (Participants) | 1
  Week 4, n=1 | 3.8100 (NA) — Standard deviation could not be calculated when number of participants was <=1

26. Other Pre Specified Outcome: Variance of HRV While Active (LF/HF)
Description: Variance of Heart Rate Variability (HRV) averaged over 5 windows of subjects being active at each protocol time point (LF/HF analysis). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data could not be calculated as participant number was <=1
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0, n=2: number analyzed (Participants) | 2
  Week 0, n=2 | 0.0000 (0.0000)
  Week 4, n=1: number analyzed (Participants) | 1
  Week 4, n=1 | 0.0000 (NA) — NA indicates that data could not be calculated as participant number was <=1

27. Other Pre Specified Outcome: Effect of Being Upright on HRV- Mean HRV (LF/HF Analysis)
Description: The effect of being upright on mean HRV was calculated as [mean HRV while sedentary not lying minus mean HRV while lying] (LF/HF analysis). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0, n=20: number analyzed (Participants) | 20
  Week 0, n=20 | 1.0563 (2.12227)
  Week 4, n=18: number analyzed (Participants) | 18
  Week 4, n=18 | 1.3507 (2.56807)
  Week 8, n=13: number analyzed (Participants) | 13
  Week 8, n=13 | 1.1937 (2.40299)
  Week 12, n=14: number analyzed (Participants) | 14
  Week 12, n=14 | 2.1585 (2.80355)
  Week 16, n=11: number analyzed (Participants) | 11
  Week 16, n=11 | 2.5080 (3.40632)
  Week 20, n=10: number analyzed (Participants) | 10
  Week 20, n=10 | 2.4613 (3.64555)
  Week 24, n=10: number analyzed (Participants) | 10
  Week 24, n=10 | 2.5161 (1.95702)
  Week 28, n=9: number analyzed (Participants) | 9
  Week 28, n=9 | -0.1964 (6.11226)
  Week 32, n=9: number analyzed (Participants) | 9
  Week 32, n=9 | 3.3476 (5.59881)
  Week 36, n=9: number analyzed (Participants) | 9
  Week 36, n=9 | 2.5583 (3.74969)
  Week 40, n=9: number analyzed (Participants) | 9
  Week 40, n=9 | 0.9722 (1.73768)
  Week 44, n=9: number analyzed (Participants) | 9
  Week 44, n=9 | 1.6069 (2.71641)
  Week 48, n=6: number analyzed (Participants) | 6
  Week 48, n=6 | 1.5796 (3.73597)

28. Other Pre Specified Outcome: Effect of Being Upright on HRV Variance (LF/HF Analysis)
Description: The effect of being upright on HRV variance was calculated as [HRV variance while sedentary not lying minus HRV variance while lying] (LF/HF analysis). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0, n=20: number analyzed (Participants) | 20
  Week 0, n=20 | -0.0750 (5.21420)
  Week 4, n=18: number analyzed (Participants) | 18
  Week 4, n=18 | -5.5005 (28.71903)
  Week 8, n=13: number analyzed (Participants) | 13
  Week 8, n=13 | -2.0885 (9.89872)
  Week 12, n=14: number analyzed (Participants) | 14
  Week 12, n=14 | 4.1473 (8.03699)
  Week 16, n=11: number analyzed (Participants) | 11
  Week 16, n=11 | 9.8909 (21.83721)
  Week 20, n=10: number analyzed (Participants) | 10
  Week 20, n=10 | 2.9204 (17.31637)
  Week 24, n=10: number analyzed (Participants) | 10
  Week 24, n=10 | -1.1979 (2.96892)
  Week 28, n=9: number analyzed (Participants) | 9
  Week 28, n=9 | -13.6310 (45.52591)
  Week 32, n=9: number analyzed (Participants) | 9
  Week 32, n=9 | -8.9054 (19.69942)
  Week 36, n=9: number analyzed (Participants) | 9
  Week 36, n=9 | 10.3525 (35.50938)
  Week 40, n=9: number analyzed (Participants) | 9
  Week 40, n=9 | -3.8092 (8.66934)
  Week 44, n=9: number analyzed (Participants) | 9
  Week 44, n=9 | -2.1221 (11.81571)
  Week 48, n=6: number analyzed (Participants) | 6
  Week 48, n=6 | 4.3165 (16.66785)

29. Other Pre Specified Outcome: Effect of Activity on Mean HRV (LF/HF)
Description: The effect of activity on mean HRV was calculated as [mean HRV while sedentary not lying minus mean HRV while lying] (LF/HF analysis). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data could not be calculated as participant number was <=1.
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0; n= 2: number analyzed (Participants) | 2
  Week 0; n= 2 | -1.6117 (2.88735)
  Week 4; n= 1: number analyzed (Participants) | 1
  Week 4; n= 1 | 0.9367 (NA) — NA indicates that data could not be calculated as participant number was <=1.

30. Other Pre Specified Outcome: Effect of Activity on HRV Variance (LF/HF Analysis)
Description: The effect of activity on HRV variance was calculated as [HRV variance while sedentary not lying minus HRV variance while lying] (LF/HF analysis). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data could not be calculated as participant number was <=1.
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Week 0; n= 2: number analyzed (Participants) | 2
  Week 0; n= 2 | -8.6500 (5.93027)
  Week 4; n= 1: number analyzed (Participants) | 1
  Week 4; n= 1 | -3.4367 (NA) — NA indicates that data could not be calculated as participant number was <=1.

31. Other Pre Specified Outcome: Mean HRV Over 24 Hours - Mean Root Mean Square of the Successive Differences (RMSSD)
Description: Mean HRV over 24 hours (RMSSD analysis), averaged for each protocol time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Milliseconds^2
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Milliseconds^2
  Week 0, n=24: number analyzed (Participants) | 24
  Week 0, n=24 | 21.2445 (6.13882)
  Week 4, n=21: number analyzed (Participants) | 21
  Week 4, n=21 | 20.0394 (6.61338)
  Week 8, n=15: number analyzed (Participants) | 15
  Week 8, n=15 | 22.4551 (5.98867)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 20.6744 (6.95469)
  Week 16, n=12: number analyzed (Participants) | 12
  Week 16, n=12 | 20.7926 (7.01048)
  Week 20, n=12: number analyzed (Participants) | 12
  Week 20, n=12 | 20.7321 (6.80432)
  Week 24, n=12: number analyzed (Participants) | 12
  Week 24, n=12 | 21.3250 (6.92749)
  Week 28, n=10: number analyzed (Participants) | 10
  Week 28, n=10 | 21.7888 (7.14731)
  Week 32, n=10: number analyzed (Participants) | 10
  Week 32, n=10 | 21.1318 (8.08213)
  Week 36, n=11: number analyzed (Participants) | 11
  Week 36, n=11 | 20.8849 (5.72665)
  Week 40, n=11: number analyzed (Participants) | 11
  Week 40, n=11 | 20.0684 (7.98572)
  Week 44, n=11: number analyzed (Participants) | 11
  Week 44, n=11 | 20.2980 (5.95832)
  Week 48, n=12: number analyzed (Participants) | 12
  Week 48, n=12 | 19.5152 (8.04882)

32. Other Pre Specified Outcome: HRV Variance Over 24 Hours - Mean Root Mean Square of the Successive Differences (RMSSD) Analysis
Description: HRV variance over 24 hours (RMSSD analysis), averaged for each protocol time point. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Milliseconds^2
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Milliseconds^2
  Week 0, n=24: number analyzed (Participants) | 24
  Week 0, n=24 | 35.3316 (25.70628)
  Week 4, n=21: number analyzed (Participants) | 21
  Week 4, n=21 | 26.2719 (19.19169)
  Week 8, n=15: number analyzed (Participants) | 15
  Week 8, n=15 | 34.5477 (18.01341)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 31.8929 (28.36635)
  Week 16, n=12: number analyzed (Participants) | 12
  Week 16, n=12 | 34.8321 (25.62477)
  Week 20, n=12: number analyzed (Participants) | 12
  Week 20, n=12 | 41.4669 (36.88159)
  Week 24, n=12: number analyzed (Participants) | 12
  Week 24, n=12 | 34.3781 (38.27469)
  Week 28, n=10: number analyzed (Participants) | 10
  Week 28, n=10 | 45.4243 (62.35269)
  Week 32, n=10: number analyzed (Participants) | 10
  Week 32, n=10 | 30.5288 (24.91715)
  Week 36, n=11: number analyzed (Participants) | 11
  Week 36, n=11 | 24.8373 (14.41668)
  Week 40, n=11: number analyzed (Participants) | 11
  Week 40, n=11 | 18.4227 (9.54924)
  Week 44, n=11: number analyzed (Participants) | 11
  Week 44, n=11 | 22.5279 (10.78475)
  Week 48, n=12: number analyzed (Participants) | 12
  Week 48, n=12 | 15.7176 (13.15760)

33. Other Pre Specified Outcome: Relationship Between Absolute Values of HRV Endpoints (LF/HF) and Absolute Value of Total ALSFRS-R
Description: Estimates for between and within subject correlation coefficients were produced following multiple linear regression analyses on the actigraphy endpoints, comparing them with the ALSFRS-R total score and the gross motor domain and fine motor domain scores. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that sample size was insufficient to calculate correlation coefficient
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Mean HRV effect of being upright v/s ALSFRS-R;n=24: number analyzed (Participants) | 24
  Mean HRV effect of being upright v/s ALSFRS-R;n=24 | 0.139
  Mean LF/HF (lying down) (1) v/s ALSFRS-R;n=25 | 0.228
  Mean LF/HF sedentary (not lying) v/s ALSFRS-R;n=24: number analyzed (Participants) | 24
  Mean LF/HF sedentary (not lying) v/s ALSFRS-R;n=24 | 0.023
  Var. LF/HF sedentary (not lying) v/s ALSFR-R;n=24: number analyzed (Participants) | 24
  Var. LF/HF sedentary (not lying) v/s ALSFR-R;n=24 | -0.041
  Mean HRV effect of activity v/s ALSFRS-R;n=3: number analyzed (Participants) | 3
  Mean HRV effect of activity v/s ALSFRS-R;n=3 | 0.421
  Mean LF/HF (avg-daytime activity) v/s ALSFRS-R;n=3: number analyzed (Participants) | 3
  Mean LF/HF (avg-daytime activity) v/s ALSFRS-R;n=3 | -0.921
  Var of HRV effect of activity v/s ALSFRS-R;n=3: number analyzed (Participants) | 3
  Var of HRV effect of activity v/s ALSFRS-R;n=3 | 0.419
  Var of HRV effect being upright v/s ALSFRS-R;n=24: number analyzed (Participants) | 24
  Var of HRV effect being upright v/s ALSFRS-R;n=24 | 0.308
  Var of LF/HF (lying down) v/s ALSFRS-R;n=25 | -0.378
  Var of LF/HF v/s ALSFRS-R;n=3: number analyzed (Participants) | 3
  Var of LF/HF v/s ALSFRS-R;n=3 | NA — NA indicates that sample size is insufficient to calculate the correlation coefficient

34. Other Pre Specified Outcome: Measurement of Speech Quality
Description: Speech quality was assessed by Central Tendency of Fundamental Frequency (CTF) F0, jitter, and shimmer for 'short ah' and 'long ah' tests. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Hertz
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Hertz
  CTF F0;Week0;n=25 (Short ah) | 151.829 (44.5983)
  CTF F0;Week12;n=18 (Short ah): number analyzed (Participants) | 18
  CTF F0;Week12;n=18 (Short ah) | 156.506 (42.0801)
  CTF F0;Week24;n=17 (Short ah): number analyzed (Participants) | 17
  CTF F0;Week24;n=17 (Short ah) | 143.481 (43.8646)
  CTF F0;Week36;n=15 (Short ah): number analyzed (Participants) | 15
  CTF F0;Week36;n=15 (Short ah) | 151.192 (43.1685)
  CTF F0;Week48;n=18 (Short ah): number analyzed (Participants) | 18
  CTF F0;Week48;n=18 (Short ah) | 156.418 (71.9125)
  CTF F0;EWD;n=3 (Short ah): number analyzed (Participants) | 3
  CTF F0;EWD;n=3 (Short ah) | 176.229 (76.2851)
  Jitter;Week0;n=25 (Short ah) | 0.405 (0.2814)
  Jitter;Week12;n=18 (Short ah): number analyzed (Participants) | 18
  Jitter;Week12;n=18 (Short ah) | 0.531 (0.2956)
  Jitter;Week24;n=17 (Short ah): number analyzed (Participants) | 17
  Jitter;Week24;n=17 (Short ah) | 0.415 (0.3345)
  Jitter;Week36;n=15 (Short ah): number analyzed (Participants) | 15
  Jitter;Week36;n=15 (Short ah) | 0.429 (0.2987)
  Jitter;Week48;n=18 (Short ah): number analyzed (Participants) | 18
  Jitter;Week48;n=18 (Short ah) | 0.379 (0.2949)
  Jitter;EWD;n=2 (Short ah): number analyzed (Participants) | 2
  Jitter;EWD;n=2 (Short ah) | 0.435 (0.1835)
  Shimmer;Week0;n=25 (Short ah) | 5.099 (1.0892)
  Shimmer;Week12;n=18 (Short ah): number analyzed (Participants) | 18
  Shimmer;Week12;n=18 (Short ah) | 5.031 (1.0850)
  Shimmer;Week24;n=17 (Short ah): number analyzed (Participants) | 17
  Shimmer;Week24;n=17 (Short ah) | 5.498 (1.1896)
  Shimmer;Week36;n=15 (Short ah): number analyzed (Participants) | 15
  Shimmer;Week36;n=15 (Short ah) | 5.203 (1.4083)
  Shimmer;Week48;n=18 (Short ah): number analyzed (Participants) | 18
  Shimmer;Week48;n=18 (Short ah) | 5.157 (1.9564)
  Shimmer;EWD;n=2 (Short ah): number analyzed (Participants) | 2
  Shimmer;EWD;n=2 (Short ah) | 5.624 (1.5979)
  CTF F0;Week0;n=25 (Long ah) | 134.443 (33.2237)
  CTF F0;Week12;n=18 (Long ah): number analyzed (Participants) | 18
  CTF F0;Week12;n=18 (Long ah) | 122.620 (35.6641)
  CTF F0;Week24;n=17 (Long ah): number analyzed (Participants) | 17
  CTF F0;Week24;n=17 (Long ah) | 146.295 (63.0013)
  CTF F0;Week36;n=15 (Long ah): number analyzed (Participants) | 15
  CTF F0;Week36;n=15 (Long ah) | 145.575 (45.5629)
  CTF F0;Week48;n=18 (Long ah): number analyzed (Participants) | 18
  CTF F0;Week48;n=18 (Long ah) | 134.198 (48.3046)
  CTF F0;EWD;n=3 (Long ah): number analyzed (Participants) | 3
  CTF F0;EWD;n=3 (Long ah) | 179.844 (25.7371)
  Jitter;Week0;n=25 (Long ah) | 0.148 (0.1701)
  Jitter;Week12;n=18 (Long ah): number analyzed (Participants) | 18
  Jitter;Week12;n=18 (Long ah) | 0.098 (0.0697)
  Jitter;Week24;n=17 (Long ah): number analyzed (Participants) | 17
  Jitter;Week24;n=17 (Long ah) | 0.178 (0.3030)
  Jitter;Week36;n=15 (Long ah): number analyzed (Participants) | 15
  Jitter;Week36;n=15 (Long ah) | 0.229 (0.3069)
  Jitter;Week48;n=18 (Long ah): number analyzed (Participants) | 18
  Jitter;Week48;n=18 (Long ah) | 0.148 (0.1309)
  Jitter;EWD;n=2 (Long ah): number analyzed (Participants) | 2
  Jitter;EWD;n=2 (Long ah) | 0.304 (0.3115)
  Shimmer;Week0;n=25 (Long ah) | 2.926 (1.0166)
  Shimmer;Week12;n=18 (Long ah): number analyzed (Participants) | 18
  Shimmer;Week12;n=18 (Long ah) | 3.192 (0.8599)
  Shimmer;Week24;n=17 (Long ah): number analyzed (Participants) | 17
  Shimmer;Week24;n=17 (Long ah) | 3.082 (1.1959)
  Shimmer;Week36;n=15 (Long ah): number analyzed (Participants) | 15
  Shimmer;Week36;n=15 (Long ah) | 2.872 (1.2162)
  Shimmer;Week48;n=18 (Long ah): number analyzed (Participants) | 18
  Shimmer;Week48;n=18 (Long ah) | 3.046 (1.4476)
  Shimmer;EWD;n=2 (Long ah): number analyzed (Participants) | 2
  Shimmer;EWD;n=2 (Long ah) | 2.767 (0.0709)

35. Other Pre Specified Outcome: Duration of Maximum Gap Between Words
Description: Duration of maximum gap between words during running speech to planned to analyze quality of speech however; was not performed.
Time Frame: Up to Week 48
Population: Full Analysis Set
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 0

36. Other Pre Specified Outcome: Speaking Rate
Description: Speaking rate was analyzed during running speech. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Words per minute
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Words per minute
  Week0; n=25 | 151.490 (42.3137)
  Week12; n=18: number analyzed (Participants) | 18
  Week12; n=18 | 160.628 (46.2482)
  Week24; n=17: number analyzed (Participants) | 17
  Week24; n=17 | 153.958 (45.2931)
  Week36; n=15: number analyzed (Participants) | 15
  Week36; n=15 | 166.342 (67.6138)
  Week48; n=18: number analyzed (Participants) | 18
  Week48; n=18 | 138.984 (65.6871)
  EWD; n=2: number analyzed (Participants) | 2
  EWD; n=2 | 179.687 (27.6064)

37. Other Pre Specified Outcome: Average Phoneme Rate
Description: Phoneme rate was analyzed for the single word "doily". Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Hertz per second
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Hertz per second
  Week0; n=25 | 6176.377 (2196.778)
  Week12; n=18: number analyzed (Participants) | 18
  Week12; n=18 | 6903.574 (2484.952)
  Week24; n=17: number analyzed (Participants) | 17
  Week24; n=17 | 5859.531 (3433.272)
  Week36; n=15: number analyzed (Participants) | 15
  Week36; n=15 | 6937.497 (4868.936)
  Week48; n=18: number analyzed (Participants) | 18
  Week48; n=18 | 5738.519 (3410.358)
  EWD; n=2: number analyzed (Participants) | 2
  EWD; n=2 | 8980.240 (709.4459)

38. Other Pre Specified Outcome: Maximum Phonation Time
Description: Maximum phonation time for the single word "doily" test was analyzed for quality of speech testing. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Seconds
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Seconds
  Week0; n=25 | 0.174 (0.0724)
  Week12; n=18: number analyzed (Participants) | 18
  Week12; n=18 | 0.188 (0.0862)
  Week24; n=17: number analyzed (Participants) | 17
  Week24; n=17 | 0.186 (0.1005)
  Week36; n=15: number analyzed (Participants) | 15
  Week36; n=15 | 0.154 (0.0608)
  Week48; n=18: number analyzed (Participants) | 18
  Week48; n=18 | 0.147 (0.0884)
  EWD; n=2: number analyzed (Participants) | 2
  EWD; n=2 | 0.212 (0.0639)

39. Other Pre Specified Outcome: Percentage Pause Time
Description: Percentage pause time for running speech was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Percentage of time
  Week0; n=25 | 31.900 (17.1724)
  Week12; n=18: number analyzed (Participants) | 18
  Week12; n=18 | 26.609 (8.1333)
  Week24; n=17: number analyzed (Participants) | 17
  Week24; n=17 | 30.177 (14.3137)
  Week36; n=15: number analyzed (Participants) | 15
  Week36; n=15 | 24.410 (9.5753)
  Week48; n=18: number analyzed (Participants) | 18
  Week48; n=18 | 23.991 (11.8426)
  EWD; n=2: number analyzed (Participants) | 2
  EWD; n=2 | 24.042 (0.3466)

40. Other Pre Specified Outcome: Relationship Between Absolute Values of Speech Endpoints and Absolute Value of ALSFRS-R
Description: Mixed Model was used to calculate Repeated Measures Correlation Coefficients between the two variables when model is converged. The correlation coefficient among the repeated measurements is same for different variables. Multiple Linear Regression was used to calculate Within and Between Participant Correlation Coefficients when Mixed Model is not converged. Data for Repeated Measures Correlation Coefficient has been presented in the table below
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  Jitter (%) (Short ah) v/s ALSFRS-R | 0.137
  CTF F0 (Long ah) v/s ALSFRS-R | -0.154
  Jitter (%) (Long ah) v/s ALSFRS-R | 0.119
  Shimmer(%) (Long ah) v/s ALSFRS-R | 0.138
  Maximum Phonation Time v/s ALSFRS-R | 0.152

41. Other Pre Specified Outcome: Relationship Between Absolute Values of Speech Endpoints and Absolute Values of FVC
Description: Mixed Model was used to calculate Repeated Measures Correlation Coefficients between the two variables when model is converged. The correlation coefficient among the repeated measurements is same for different variables. Multiple Linear Regression was used to calculate Within and Between Participant Correlation Coefficients when Mixed Model is not converged. Data for Between Subject Correlation Coefficient has been presented in the table below
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Ratio
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Ratio
  CTF F0 (Short ah) v/s FVC | -0.214
  Jitter (%) (Short ah) v/s FVC | 0.143
  Shimmer(%) (Short ah) v/s FVC | -0.080
  CTF F0 (Long ah) v/s FVC | -0.504
  Jitter (%) (Long ah) v/s FVC | -0.321
  Shimmer(%) (Long ah) v/s FVC | -0.327
  Average Phoneme Rate v/s FVC | 0.453
  Maximum Phonation Time v/s FVC | -0.215
  Percent Pause Time v/s FVC | -0.376
  Speaking Rate v/s FVC | 0.547

42. Other Pre Specified Outcome: Number of Participants Reporting Sensor Comfort
Description: Participant's feedback on whether the sensor was comfortable to wear was categorized as "yes" and "no". Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Participants
  Sensor comfortable to wear;Pilot; n=5;Yes: number analyzed (Participants) | 5
  Sensor comfortable to wear;Pilot; n=5;Yes | 4
  Sensor comfortable to wear;Pilot; n=5;No: number analyzed (Participants) | 5
  Sensor comfortable to wear;Pilot; n=5;No | 1
  Sensor comfortable to wear;Pilot repeat; n=5;Yes: number analyzed (Participants) | 5
  Sensor comfortable to wear;Pilot repeat; n=5;Yes | 3
  Sensor comfortable to wear;Pilot repeat; n=5;No: number analyzed (Participants) | 5
  Sensor comfortable to wear;Pilot repeat; n=5;No | 2
  Sensor comfortable to wear;Week12; n=15;Yes: number analyzed (Participants) | 15
  Sensor comfortable to wear;Week12; n=15;Yes | 14
  Sensor comfortable to wear;Week12; n=15;No: number analyzed (Participants) | 15
  Sensor comfortable to wear;Week12; n=15;No | 1
  Sensor comfortable to wear;Week24; n=14; Yes: number analyzed (Participants) | 14
  Sensor comfortable to wear;Week24; n=14; Yes | 13
  Sensor comfortable to wear;Week24; n=14;No: number analyzed (Participants) | 14
  Sensor comfortable to wear;Week24; n=14;No | 1
  Sensor comfortable to wear;Week36; n=14; Yes: number analyzed (Participants) | 14
  Sensor comfortable to wear;Week36; n=14; Yes | 12
  Sensor comfortable to wear;Week36; n=14; No: number analyzed (Participants) | 14
  Sensor comfortable to wear;Week36; n=14; No | 2
  Sensor comfortable to wear;Week48; n=18; Yes: number analyzed (Participants) | 18
  Sensor comfortable to wear;Week48; n=18; Yes | 14
  Sensor comfortable to wear;Week48; n=18;No: number analyzed (Participants) | 18
  Sensor comfortable to wear;Week48; n=18;No | 4
  Sensor comfortable to wear;EWD; n=2;Yes: number analyzed (Participants) | 2
  Sensor comfortable to wear;EWD; n=2;Yes | 0
  Sensor comfortable to wear;EWD; n=2;No: number analyzed (Participants) | 2
  Sensor comfortable to wear;EWD; n=2;No | 2

43. Other Pre Specified Outcome: Number of Participants Reporting Impact on Sleep
Description: Participant feedback on how much the sensor impacted their sleep was categorized as "not at all", "moderately" and "minimally". Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Participants
  Not at all;Pilot; n=5: number analyzed (Participants) | 5
  Not at all;Pilot; n=5 | 4
  Moderately;Pilot; n=5: number analyzed (Participants) | 5
  Moderately;Pilot; n=5 | 1
  Minimally; Pilot; n=5: number analyzed (Participants) | 5
  Minimally; Pilot; n=5 | 0
  Not at all;Pilot repeat; n=5: number analyzed (Participants) | 5
  Not at all;Pilot repeat; n=5 | 3
  Moderately;Pilot repeat; n=5: number analyzed (Participants) | 5
  Moderately;Pilot repeat; n=5 | 2
  Minimally; Pilot repeat; n=5: number analyzed (Participants) | 5
  Minimally; Pilot repeat; n=5 | 0
  Not at all;Week12; n=15: number analyzed (Participants) | 15
  Not at all;Week12; n=15 | 15
  Moderately;Week12; n=15: number analyzed (Participants) | 15
  Moderately;Week12; n=15 | 0
  Minimally; Week12; n=15: number analyzed (Participants) | 15
  Minimally; Week12; n=15 | 0
  Not at all;Week24; n=14: number analyzed (Participants) | 14
  Not at all;Week24; n=14 | 12
  Moderately;Week24; n=14: number analyzed (Participants) | 14
  Moderately;Week24; n=14 | 0
  Minimally; Week24; n=14: number analyzed (Participants) | 14
  Minimally; Week24; n=14 | 2
  Not at all;Week36; n=14: number analyzed (Participants) | 14
  Not at all;Week36; n=14 | 12
  Moderately;Week36; n=14: number analyzed (Participants) | 14
  Moderately;Week36; n=14 | 0
  Minimally; Week36; n=14: number analyzed (Participants) | 14
  Minimally; Week36; n=14 | 2
  Not at all;Week48; n=18: number analyzed (Participants) | 18
  Not at all;Week48; n=18 | 15
  Moderately;Week48; n=18: number analyzed (Participants) | 18
  Moderately;Week48; n=18 | 0
  Minimally; Week48; n=18: number analyzed (Participants) | 18
  Minimally; Week48; n=18 | 3
  Not at all;EWD; n=2: number analyzed (Participants) | 2
  Not at all;EWD; n=2 | 1
  Moderately;EWD; n=2: number analyzed (Participants) | 2
  Moderately;EWD; n=2 | 1
  Minimally; EWD; n=2: number analyzed (Participants) | 2
  Minimally; EWD; n=2 | 0

44. Other Pre Specified Outcome: Number of Participants With Ease of Setting up and Attaching the Sensor
Description: The participants were required to give feedback on how easy was it to set up and/ or attach the sensor and it was categorized as "easy", "neutral" and "difficult". Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Participants
  Easy;Pilot; n=5: number analyzed (Participants) | 5
  Easy;Pilot; n=5 | 4
  Neutral;Pilot; n=5: number analyzed (Participants) | 5
  Neutral;Pilot; n=5 | 1
  Difficult;Pilot; n=5: number analyzed (Participants) | 5
  Difficult;Pilot; n=5 | 0
  Easy;Pilot repeat; n=5: number analyzed (Participants) | 5
  Easy;Pilot repeat; n=5 | 5
  Neutral;Pilot repeat; n=5: number analyzed (Participants) | 5
  Neutral;Pilot repeat; n=5 | 0
  Difficult;Pilot repeat; n=5: number analyzed (Participants) | 5
  Difficult;Pilot repeat; n=5 | 0
  Easy;Week0; n=25 | 23
  Neutral;Week0; n=25 | 2
  Difficult;Week0; n=25 | 0
  Easy;Week4; n=23: number analyzed (Participants) | 23
  Easy;Week4; n=23 | 23
  Neutral;Week4; n=23: number analyzed (Participants) | 23
  Neutral;Week4; n=23 | 0
  Difficult;Week4; n=23: number analyzed (Participants) | 23
  Difficult;Week4; n=23 | 0
  Easy;Week8; n=21: number analyzed (Participants) | 21
  Easy;Week8; n=21 | 19
  Neutral;Week8; n=21: number analyzed (Participants) | 21
  Neutral;Week8; n=21 | 0
  Difficult;Week8; n=21: number analyzed (Participants) | 21
  Difficult;Week8; n=21 | 2
  Easy;Week12; n=20: number analyzed (Participants) | 20
  Easy;Week12; n=20 | 18
  Neutral;Week12; n=20: number analyzed (Participants) | 20
  Neutral;Week12; n=20 | 2
  Difficult;Week12; n=20: number analyzed (Participants) | 20
  Difficult;Week12; n=20 | 0
  Easy;Week16; n=18: number analyzed (Participants) | 18
  Easy;Week16; n=18 | 15
  Neutral;Week16; n=18: number analyzed (Participants) | 18
  Neutral;Week16; n=18 | 2
  Difficult;Week16; n=18: number analyzed (Participants) | 18
  Difficult;Week16; n=18 | 1
  Easy;Week20; n=20: number analyzed (Participants) | 20
  Easy;Week20; n=20 | 15
  Neutral;Week20; n=20: number analyzed (Participants) | 20
  Neutral;Week20; n=20 | 2
  Difficult;Week20; n=20: number analyzed (Participants) | 20
  Difficult;Week20; n=20 | 3
  Easy;Week24; n=18: number analyzed (Participants) | 18
  Easy;Week24; n=18 | 15
  Neutral;Week24; n=18: number analyzed (Participants) | 18
  Neutral;Week24; n=18 | 2
  Difficult;Week24; n=18: number analyzed (Participants) | 18
  Difficult;Week24; n=18 | 1
  Easy;Week28; n=16: number analyzed (Participants) | 16
  Easy;Week28; n=16 | 12
  Neutral;Week28; n=16: number analyzed (Participants) | 16
  Neutral;Week28; n=16 | 2
  Difficult;Week28; n=16: number analyzed (Participants) | 16
  Difficult;Week28; n=16 | 2
  Easy;Week32; n=20: number analyzed (Participants) | 20
  Easy;Week32; n=20 | 15
  Neutral;Week32; n=20: number analyzed (Participants) | 20
  Neutral;Week32; n=20 | 3
  Difficult;Week32; n=20: number analyzed (Participants) | 20
  Difficult;Week32; n=20 | 2
  Easy;Week36; n=18: number analyzed (Participants) | 18
  Easy;Week36; n=18 | 14
  Neutral;Week36; n=18: number analyzed (Participants) | 18
  Neutral;Week36; n=18 | 3
  Difficult;Week36; n=18: number analyzed (Participants) | 18
  Difficult;Week36; n=18 | 1
  Easy;Week40; n=15: number analyzed (Participants) | 15
  Easy;Week40; n=15 | 10
  Neutral;Week40; n=15: number analyzed (Participants) | 15
  Neutral;Week40; n=15 | 3
  Difficult;Week40; n=15: number analyzed (Participants) | 15
  Difficult;Week40; n=15 | 2
  Easy;Week44; n=16: number analyzed (Participants) | 16
  Easy;Week44; n=16 | 13
  Neutral;Week44; n=16: number analyzed (Participants) | 16
  Neutral;Week44; n=16 | 1
  Difficult;Week44; n=16: number analyzed (Participants) | 16
  Difficult;Week44; n=16 | 2
  Easy;Week48; n=15: number analyzed (Participants) | 15
  Easy;Week48; n=15 | 8
  Neutral;Week48; n=15: number analyzed (Participants) | 15
  Neutral;Week48; n=15 | 3
  Difficult;Week48; n=15: number analyzed (Participants) | 15
  Difficult;Week48; n=15 | 4

45. Other Pre Specified Outcome: Number of Participants With Corresponding Activity Level Required to Complete Their Job
Description: The activity level required by the participant to complete their job was recorded, and was categorized as Not working, Physical activity required, and Sedentary. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Participants
  Pilot; Not working;n=5: number analyzed (Participants) | 5
  Pilot; Not working;n=5 | 1
  Pilot; Physical activity required;n=5: number analyzed (Participants) | 5
  Pilot; Physical activity required;n=5 | 2
  Pilot; Sedentary;n=5: number analyzed (Participants) | 5
  Pilot; Sedentary;n=5 | 2
  Pilot repeat; Not working;n=5: number analyzed (Participants) | 5
  Pilot repeat; Not working;n=5 | 1
  Pilot Repeat; Physical activity required;n=5: number analyzed (Participants) | 5
  Pilot Repeat; Physical activity required;n=5 | 0
  Pilot Repeat; Sedentary;n=5: number analyzed (Participants) | 5
  Pilot Repeat; Sedentary;n=5 | 4
  Week0; Not working;n=25 | 10
  Week0; Physical activity required;n=25 | 10
  Week0; Sedentary;n=25 | 5
  Week4; Not working;n=23: number analyzed (Participants) | 23
  Week4; Not working;n=23 | 8
  Week4; Physical activity required;n=23: number analyzed (Participants) | 23
  Week4; Physical activity required;n=23 | 7
  Week4; Sedentary;n=23: number analyzed (Participants) | 23
  Week4; Sedentary;n=23 | 8
  Week8; Not working;n=21: number analyzed (Participants) | 21
  Week8; Not working;n=21 | 12
  Week8; Physical activity required;n=21: number analyzed (Participants) | 21
  Week8; Physical activity required;n=21 | 5
  Week8; Sedentary;n=21: number analyzed (Participants) | 21
  Week8; Sedentary;n=21 | 4
  Week12; Not working;n=20: number analyzed (Participants) | 20
  Week12; Not working;n=20 | 8
  Week12; Physical activity required;n=20: number analyzed (Participants) | 20
  Week12; Physical activity required;n=20 | 5
  Week12; Sedentary;n=20: number analyzed (Participants) | 20
  Week12; Sedentary;n=20 | 7
  Week16; Not working;n=18: number analyzed (Participants) | 18
  Week16; Not working;n=18 | 11
  Week16; Physical activity required;n=18: number analyzed (Participants) | 18
  Week16; Physical activity required;n=18 | 3
  Week16; Sedentary;n=18: number analyzed (Participants) | 18
  Week16; Sedentary;n=18 | 4
  Week20; Not working;n=20: number analyzed (Participants) | 20
  Week20; Not working;n=20 | 11
  Week20; Physical activity required;n=20: number analyzed (Participants) | 20
  Week20; Physical activity required;n=20 | 5
  Week20; Sedentary;n=20: number analyzed (Participants) | 20
  Week20; Sedentary;n=20 | 4
  Week24; Not working;n=18: number analyzed (Participants) | 18
  Week24; Not working;n=18 | 11
  Week24; Physical activity required;n=18: number analyzed (Participants) | 18
  Week24; Physical activity required;n=18 | 4
  Week24; Sedentary;n=18: number analyzed (Participants) | 18
  Week24; Sedentary;n=18 | 3
  Week28; Not working;n=16: number analyzed (Participants) | 16
  Week28; Not working;n=16 | 9
  Week28; Physical activity required;n=16: number analyzed (Participants) | 16
  Week28; Physical activity required;n=16 | 2
  Week28; Sedentary;n=16: number analyzed (Participants) | 16
  Week28; Sedentary;n=16 | 5
  Week32; Not working;n=20: number analyzed (Participants) | 20
  Week32; Not working;n=20 | 11
  Week32; Physical activity required;n=20: number analyzed (Participants) | 20
  Week32; Physical activity required;n=20 | 5
  Week32; Sedentary;n=20: number analyzed (Participants) | 20
  Week32; Sedentary;n=20 | 4
  Week36; Not working;n=18: number analyzed (Participants) | 18
  Week36; Not working;n=18 | 11
  Week36; Physical activity required;n=18: number analyzed (Participants) | 18
  Week36; Physical activity required;n=18 | 3
  Week36; Sedentary;n=18: number analyzed (Participants) | 18
  Week36; Sedentary;n=18 | 4
  Week40; Not working;n=15: number analyzed (Participants) | 15
  Week40; Not working;n=15 | 7
  Week40; Physical activity required;n=15: number analyzed (Participants) | 15
  Week40; Physical activity required;n=15 | 7
  Week40; Sedentary;n=15: number analyzed (Participants) | 15
  Week40; Sedentary;n=15 | 1
  Week44; Not working;n=16: number analyzed (Participants) | 16
  Week44; Not working;n=16 | 8
  Week44; Physical activity required;n=16: number analyzed (Participants) | 16
  Week44; Physical activity required;n=16 | 4
  Week44; Sedentary;n=16: number analyzed (Participants) | 16
  Week44; Sedentary;n=16 | 4
  Week48; Not working;n=15: number analyzed (Participants) | 15
  Week48; Not working;n=15 | 7
  Week48; Physical activity required;n=15: number analyzed (Participants) | 15
  Week48; Physical activity required;n=15 | 4
  Week48; Sedentary;n=15: number analyzed (Participants) | 15
  Week48; Sedentary;n=15 | 4

46. Other Pre Specified Outcome: Number of Participants With Corresponding Average Activity Level During Time of Wearing the Sensor
Description: Average activity level during the time of wearing the sensor was reported by the participants, and was categorized as very low level activity, low level activity, moderate level activity and high level activity. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Participants
  Pilot;Very low level activity;n=5: number analyzed (Participants) | 5
  Pilot;Very low level activity;n=5 | 0
  Pilot; Low level activity; n=5: number analyzed (Participants) | 5
  Pilot; Low level activity; n=5 | 2
  Pilot;Moderate level activity;n=5: number analyzed (Participants) | 5
  Pilot;Moderate level activity;n=5 | 3
  Pilot;High level activity;n=5: number analyzed (Participants) | 5
  Pilot;High level activity;n=5 | 0
  Pilot repeat;Very low level activity;n=5: number analyzed (Participants) | 5
  Pilot repeat;Very low level activity;n=5 | 1
  Pilot repeat; Low level activity; n=5: number analyzed (Participants) | 5
  Pilot repeat; Low level activity; n=5 | 2
  Pilot repeat;Moderate level activity;n=5: number analyzed (Participants) | 5
  Pilot repeat;Moderate level activity;n=5 | 2
  Pilot repeat;High level activity;n=5: number analyzed (Participants) | 5
  Pilot repeat;High level activity;n=5 | 0
  Week0;Very low level activity;n=25 | 2
  Week0;Low level activity;n=25 | 6
  Week0;Moderate level activity;n=25 | 14
  Week0;High level activity;n=25 | 3
  Week4;Very low level activity;n=23: number analyzed (Participants) | 23
  Week4;Very low level activity;n=23 | 2
  Week4;Low level activity;n=23: number analyzed (Participants) | 23
  Week4;Low level activity;n=23 | 9
  Week4;Moderate level activity;n=23: number analyzed (Participants) | 23
  Week4;Moderate level activity;n=23 | 11
  Week4;High level activity;n=23: number analyzed (Participants) | 23
  Week4;High level activity;n=23 | 1
  Week8;Very low level activity;n=21: number analyzed (Participants) | 21
  Week8;Very low level activity;n=21 | 0
  Week8;Low level activity;n=21: number analyzed (Participants) | 21
  Week8;Low level activity;n=21 | 11
  Week8;Moderate level activity;n=21: number analyzed (Participants) | 21
  Week8;Moderate level activity;n=21 | 9
  Week8;High level activity;n=21: number analyzed (Participants) | 21
  Week8;High level activity;n=21 | 1
  Week12;Very low level activity;n=20: number analyzed (Participants) | 20
  Week12;Very low level activity;n=20 | 2
  Week12;Low level activity;n=20: number analyzed (Participants) | 20
  Week12;Low level activity;n=20 | 11
  Week12;Moderate level activity;n=20: number analyzed (Participants) | 20
  Week12;Moderate level activity;n=20 | 6
  Week12;High level activity;n=20: number analyzed (Participants) | 20
  Week12;High level activity;n=20 | 1
  Week16;Very low level activity;n=18: number analyzed (Participants) | 18
  Week16;Very low level activity;n=18 | 1
  Week16;Low level activity;n=18: number analyzed (Participants) | 18
  Week16;Low level activity;n=18 | 9
  Week16;Moderate level activity;n=18: number analyzed (Participants) | 18
  Week16;Moderate level activity;n=18 | 8
  Week16;High level activity;n=18: number analyzed (Participants) | 18
  Week16;High level activity;n=18 | 0
  Week20;Very low level activity;n=20: number analyzed (Participants) | 20
  Week20;Very low level activity;n=20 | 0
  Week20;Low level activity;n=20: number analyzed (Participants) | 20
  Week20;Low level activity;n=20 | 14
  Week20;Moderate level activity;n=20: number analyzed (Participants) | 20
  Week20;Moderate level activity;n=20 | 5
  Week20;High level activity;n=20: number analyzed (Participants) | 20
  Week20;High level activity;n=20 | 1
  Week24;Very low level activity;n=18: number analyzed (Participants) | 18
  Week24;Very low level activity;n=18 | 0
  Week24;Low level activity;n=18: number analyzed (Participants) | 18
  Week24;Low level activity;n=18 | 10
  Week24;Moderate level activity;n=18: number analyzed (Participants) | 18
  Week24;Moderate level activity;n=18 | 7
  Week24;High level activity;n=18: number analyzed (Participants) | 18
  Week24;High level activity;n=18 | 1
  Week28;Very low level activity;n=16: number analyzed (Participants) | 16
  Week28;Very low level activity;n=16 | 1
  Week28;Low level activity;n=16: number analyzed (Participants) | 16
  Week28;Low level activity;n=16 | 10
  Week28;Moderate level activity;n=16: number analyzed (Participants) | 16
  Week28;Moderate level activity;n=16 | 3
  Week28;High level activity;n=16: number analyzed (Participants) | 16
  Week28;High level activity;n=16 | 2
  Week32;Very low level activity;n=20: number analyzed (Participants) | 20
  Week32;Very low level activity;n=20 | 4
  Week32;Low level activity;n=20: number analyzed (Participants) | 20
  Week32;Low level activity;n=20 | 10
  Week32;Moderate level activity;n=20: number analyzed (Participants) | 20
  Week32;Moderate level activity;n=20 | 4
  Week32;High level activity;n=20: number analyzed (Participants) | 20
  Week32;High level activity;n=20 | 2
  Week36;Very low level activity;n=18: number analyzed (Participants) | 18
  Week36;Very low level activity;n=18 | 3
  Week36;Low level activity;n=18: number analyzed (Participants) | 18
  Week36;Low level activity;n=18 | 9
  Week36;Moderate level activity;n=18: number analyzed (Participants) | 18
  Week36;Moderate level activity;n=18 | 3
  Week36;High level activity;n=18: number analyzed (Participants) | 18
  Week36;High level activity;n=18 | 3
  Week40;Very low level activity;n=15: number analyzed (Participants) | 15
  Week40;Very low level activity;n=15 | 3
  Week40;Low level activity;n=15: number analyzed (Participants) | 15
  Week40;Low level activity;n=15 | 7
  Week40;Moderate level activity;n=15: number analyzed (Participants) | 15
  Week40;Moderate level activity;n=15 | 4
  Week40;High level activity;n=15: number analyzed (Participants) | 15
  Week40;High level activity;n=15 | 1
  Week44;Very low level activity;n=16: number analyzed (Participants) | 16
  Week44;Very low level activity;n=16 | 2
  Week44;Low level activity;n=16: number analyzed (Participants) | 16
  Week44;Low level activity;n=16 | 8
  Week44;Moderate level activity;n=16: number analyzed (Participants) | 16
  Week44;Moderate level activity;n=16 | 6
  Week44;High level activity;n=16: number analyzed (Participants) | 16
  Week44;High level activity;n=16 | 0
  Week48;Very low level activity;n=15: number analyzed (Participants) | 15
  Week48;Very low level activity;n=15 | 2
  Week48;Low level activity;n=15: number analyzed (Participants) | 15
  Week48;Low level activity;n=15 | 7
  Week48;Moderate level activity;n=15: number analyzed (Participants) | 15
  Week48;Moderate level activity;n=15 | 5
  Week48;High level activity;n=15: number analyzed (Participants) | 15
  Week48;High level activity;n=15 | 1

47. Other Pre Specified Outcome: Number of Participants Whose Sensor Fell Off
Description: The participants reported whether the sensor fell off. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 48
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Participants
  Pilot;Yes;n=5: number analyzed (Participants) | 5
  Pilot;Yes;n=5 | 0
  Pilot;No;n=5: number analyzed (Participants) | 5
  Pilot;No;n=5 | 5
  Pilot Repeat;Yes;n=5: number analyzed (Participants) | 5
  Pilot Repeat;Yes;n=5 | 1
  Pilot Repeat;No;n=5: number analyzed (Participants) | 5
  Pilot Repeat;No;n=5 | 4
  Week 0; Yes; n=25 | 0
  Week 0; No; n=25 | 25
  Week 4; Yes;n=23: number analyzed (Participants) | 23
  Week 4; Yes;n=23 | 2
  Week 4;No; n=23: number analyzed (Participants) | 23
  Week 4;No; n=23 | 21
  Week 8; Yes; n=21: number analyzed (Participants) | 21
  Week 8; Yes; n=21 | 4
  Week 8; No; n=21: number analyzed (Participants) | 21
  Week 8; No; n=21 | 17
  Week 12; Yes;n=20: number analyzed (Participants) | 20
  Week 12; Yes;n=20 | 1
  Week 12;No;n=20: number analyzed (Participants) | 20
  Week 12;No;n=20 | 19
  Week 16;Yes; n=18: number analyzed (Participants) | 18
  Week 16;Yes; n=18 | 0
  Week 16;No; n=18: number analyzed (Participants) | 18
  Week 16;No; n=18 | 18
  Week 20; Yes; n=20: number analyzed (Participants) | 20
  Week 20; Yes; n=20 | 1
  Week 20; No; n=20: number analyzed (Participants) | 20
  Week 20; No; n=20 | 19
  Week 24;Yes; n=18: number analyzed (Participants) | 18
  Week 24;Yes; n=18 | 2
  Week 24;No; n=18: number analyzed (Participants) | 18
  Week 24;No; n=18 | 16
  Week 28;Yes; n=16: number analyzed (Participants) | 16
  Week 28;Yes; n=16 | 1
  Week 28;No; n=16: number analyzed (Participants) | 16
  Week 28;No; n=16 | 15
  Week 32;Yes; n=20: number analyzed (Participants) | 20
  Week 32;Yes; n=20 | 1
  Week 32;No; n=20: number analyzed (Participants) | 20
  Week 32;No; n=20 | 19
  Week 36;Yes; n=18: number analyzed (Participants) | 18
  Week 36;Yes; n=18 | 0
  Week 36;No; n=18: number analyzed (Participants) | 18
  Week 36;No; n=18 | 18
  Week 40;Yes; n=15: number analyzed (Participants) | 15
  Week 40;Yes; n=15 | 1
  Week 40;No; n=15: number analyzed (Participants) | 15
  Week 40;No; n=15 | 14
  Week 44;Yes; n=16: number analyzed (Participants) | 16
  Week 44;Yes; n=16 | 0
  Week 44;No; n=16: number analyzed (Participants) | 16
  Week 44;No; n=16 | 16
  Week 48;Yes; n=15: number analyzed (Participants) | 15
  Week 48;Yes; n=15 | 0
  Week 48;No; n=15: number analyzed (Participants) | 15
  Week 48;No; n=15 | 15

48. Other Pre Specified Outcome: Number of Participants With Adverse Events Secondary to the Devices Used or Due to Study Procedures
Description: Only those AEs and SAEs which, in the opinion of the investigator, were related to a protocol-mandated procedure or one of the devices used in the study were reported. An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or event associated with liver injury and impaired liver function were categorized as SAE.
Time Frame: Up to Week 48
Population: Safety Population comprised of all participants who carried out at least one protocol specified procedure
Measure: Number; unit: Participants
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Participants
  AEs | 6
  SAEs | 0

49. Other Pre Specified Outcome: Type of Adverse Events Secondary to the Devices Used or Due to Study Procedures
Description: Only those AEs and SAEs which, in the opinion of the investigator, were related to a protocol-mandated procedure or one of the devices used in the study were reported. An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or event associated with liver injury and impaired liver function were categorized as SAE. Number of AEs, SAEs and Adverse events leading to discontinuation (AELDs)from the study is presented
Time Frame: Up to Week 48
Population: Safety Population
Measure: Number; unit: Events
Arm/Group | Mega Faros Device + Fast Fix
Number analyzed (Participants) | 25
Events
  AEs | 6
  SAEs | 0

ADVERSE EVENTS:
Time Frame: On-treatment SAEs and non-serious AEs were collected from start of study treatment until Week 48.
Description: On-treatment SAEs and non-serious AEs are reported for Safety Population
Groups:
- Mega Faros Device + Fast Fix: During Pilot phase,subjects will attend clinic at least once to perform a series of set reference tasks while wearing the accelerometer and electrode. Subjects will also continuously wear the accelerometer and electrode in their routine home-life setting for approximately 3 days after the clinic visit (home monitoring). During 48 week Core Study, subjects will attend 5 clinic visits to perform gold standard measures of function (ALS Functional Rating Scale-Revised and Forced Vital Capacity) and perform a series of set reference tasks while wearing the accelerometer and electrode. Subjects will also continuously wear the accelerometer and electrode in their routine home-life setting for approximately 3 days after the clinic visits (home monitoring). In between clinic visits, subjects will attach the accelerometer and electrode and wear it for approximately 3 days in their home. A telephone contact with the subject will be made by the site at the end of each 3-day home monitoring period
Arm/Group | Mega Faros Device + Fast Fix
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mega Faros Device + Fast Fix (N=25)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT02447952/SAP_000.pdf
  • Study Protocol (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT02447952/Prot_001.pdf